

Study report CRO-PK-20-345 Sponsor code LDX0219 Ladarixin 200 mg capsules - food effect Final version 1.0, 05OCT21

# 16.1.9 Documentation of statistical and pharmacokinetic methods

The following document is enclosed:

> Statistical analysis plan including table and listing shells, Final version 1.0, 10FEB21



# STATISTICAL ANALYSIS PLAN

Study CRO-PK-20-345 - Sponsor code LDX0219

# Influence of Food on the Oral Bioavailability of Ladarixin 200 mg Capsule in Healthy Volunteers of Both Sexes. A Single dose (400 mg), Randomized, Open Label, Two-Way Crossover Study

Single center, single dose, open label, randomized, two-way, crossover, food effect study

Test treatment Ladarixin 200 mg hard gelatin capsules, Dompé farmaceutici

(fed conditions): S.p.A., Italy

Reference treatment Ladarixin 200 mg hard gelatin capsules, Dompé farmaceutici

(fasting conditions): S.p.A., Italy

Sponsor: Dompé farmaceutici S.p.A.,

via Santa Lucia 6; 20122 Milan, Italy

Phone: +39 02.58383.1 Fax: +39 02.58383.324

Email: pieradelchi.ruffini@dompe.com

Sponsor Medical Expert:

Pier Adelchi Ruffini, MD -Global Clinical Development Director

Investigator: Milko Radicioni, MD - Principal investigator

CROSS Research S.A., Phase I Unit

Via F.A. Giorgioli 14

CH-6864 Arzo, Switzerland Phone: +41.91.64.04.450 Fax: +41.91.64.04.451

Email: clinic@croalliance.com

Development phase: Phase I

Version and date: Final version 1.0, 10FEB2021

This study will be conducted in accordance with current version of Good Clinical Practice (GCP), ICH topic E6 (R2)

Property of the sponsor

May not be used, divulged, published or otherwise disclosed without the consent of the sponsor

This document comprises 34 pages plus appendices



# **VERSIONS' HISTORY**

| Version Date of Issue | | Reason for change |
|---|---|---|
| Draft version 0.1 | 31DEC2020 | Francesca Morano issued the first draft |
| Draft version 0.2 | 15JAN2021 | Francesca Morano issue the second draft after internal revision |
| Pre-final version 0.3 | 02FEB2021 | Francesca Morano issued pre-final version 0.3 after sponsor revision |
| Final version 1.0 | 10FEB2021 | Francesca Morano issued final version 1.0 after sponsor approval |



# APPROVAL AND ACKNOWLEDGEMENT

Dompé farmaceutici S.p.A., Italy

| Sponsor Trial Manager<br>Giuseppe Terpolilli, PharmD, O | Clinical Ope | erations Specialist | |
|---|---|---|---|
| 10/02/2021 | | Mingo | The solifle |
| Date | Signature | of M | |
| <b>Sponsor Statistical Expert</b> | | | |
| Giovanni Goisis, Sponsor Princ | cipal Biosta | tistician | |
| 10/02/2021 | | Cuoven | 2016-8 |
| Date | Signature | | / |





| CRO<br>CROSS Research S.A. | |
|---|---|
| CROSS Research S.A. | |
| Statistical Analysis (for appr<br>Francesca Morano, Junior Bios | statistician and Data Manager |
| 10 FEB 2021 | France Macmo |
| Date | Signature |
| Biometry Unit Representativ<br>Alessandra Gentili, Biometry M | re (for approval and acknowledgement)<br>Manager, Unit Head |
| 10FEB 2021 | Alessona fel ' |
| Date | Signature |
| Andrea Di Stefano, Senior Med | adread Stope |
| Date | Signature |
| Chiara Leuratti, Clinical Projec | entative (for acknowledgement only) ets Unit Head |
| NOTER WY | Signature |
| Daic | Signature |



# STUDY SCHEDULE

| ACTIVITIES | Scree | ning | | PERIOI | ) 1 | (wash- | | PER | IOD 2 | | Final visit/ETV <sup>1</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit | V1 | V1.1 | V2 | | V3 | out≥14 days) | V4 | V5 | | V6 | Final VISIUE I V |
| | Day -21/-2 | Day -3<br>or -2 | Day -1 | Day 1 | Days 2, 3, 4 | | Day -3<br>or -2 | Day -1 | Day 1 | Days 2, 3, 4 | Day 4 of period 2 <sup>2</sup> or early termination |
| Informed consent | X | | | | | | | | | | |
| Demography | X | | | | | | | | | | |
| Lifestyle | X | | | | | | | | | | |
| Medical history and underlying disease | x | | | | | | | | | | |
| Physical abnormalities | X | | | | x <sup>3</sup> | | | х | | | X |
| Previous and concomitant medications | x | х | X | X | x | х | Х | x | X | X | x |
| Height and Body Mass Index | X | | | | | | | | | | |
| Body Weight | X | | | | x <sup>3</sup> | | | х | | | X |
| Laboratory analysis <sup>4</sup> | X | | | | | | | | | | X |
| Virology | X | | | | | | | | | | |
| SARS-COV2 test | | X | | | | | X | | | | |
| Pregnancy test | x <sup>5</sup> | | $\mathbf{x}^6$ | | | | | x <sup>6</sup> | | | x <sup>5</sup> |
| Urine drug screening <sup>7</sup> | X | | X | | | | | X | | | X |
| Alcohol breath test | X | | X | | | | | X | | | X |
| Coagulation | X | | | | | | | | | | |
| Vital signs <sup>10</sup> | X | | X | x <sup>8</sup> | x <sup>9</sup> | | | X | x <sup>8</sup> | $x^9$ | x <sup>11</sup> |
| ECG | X | | X | x <sup>8</sup> | x <sup>9</sup> | | | X | x <sup>8</sup> | x <sup>9</sup> | x <sup>11</sup> |
| Inclusion/exclusion criteria | X | | X | | | | | X | | | |
| Subject eligibility | X | | X | | | | | X | | | |
| Enrolment / randomization | | | X | | | | | | | | |
| Confinement | | | X | X | X | | | X | X | X | |
| Discharge | | | | | x <sup>12</sup> | | | | 12 | | X |
| Study dosing | | | | x <sup>13</sup> | | | | | x <sup>13</sup> | | |
| Blood samplings | | | | x <sup>14</sup> | x <sup>14</sup> | | | | x <sup>14</sup> | x <sup>14</sup> | |
| Standardized meals | | | x <sup>15</sup> | x <sup>16</sup> | x <sup>17</sup> | | | x <sup>15</sup> | x <sup>16</sup> | x <sup>17</sup> | |
| Adverse events monitoring <sup>18</sup> | X | X | X | X | X | X | X | X | X | X | X |

CROSS Research S.A.




Statistical analysis plan CRO-PK-20-345 Sponsor code LDX0219 Ladarixin 200 mg capsules - food effect Final version 1.0, 10FEB2021

- 1. Early termination visit (ETV) in case of premature discontinuation
- 2. Final visit on day 4 of period 2 after the 72-h post-dose blood sampling
- 3. On day 4 of period 1, upon discharge
- 4. Hematology, blood chemistry and urinalysis
- 5. Serum  $\beta$ -HCG test (women only)
- 6. Urine pregnancy test (women only)
- 7. Multi-drug kit (cocaine, amphetamine, methamphetamine, cannabinoids [△-9-tetrahydrocannabinol-THC], opiates and ecstasy)
- 8. At pre-dose
- 9. At 72 h post-dose (corresponding to the final visit assessment in period 2)
- 10. Blood pressure, heart rate, body temperature
- 11. ETV only
- 12. In the morning of day 4 of period 1
- 13. At 08:00±1 h
- 14. At pre-dose (0), 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 30, 36, 48, 54, 60 and 72 h post-dose
- 15. Standardized low-fat dinner served in the evening
- 16. Subjects allocated to the fed condition (T treatment) only: a high-fat and high-caloric breakfast to be started 30 min pre-dose and completed within 30 min. Standardized lunch and dinner at approximately 13:00 (5 h post-dose on day 1) and 20:00 (12 h post-dose on day 1) in both periods
- 17. Standardized breakfast, lunch and dinner served on days 2 and 3 at approximately 09:00, 13:00 and 20:00, respectively
- 18. Adverse events monitored starting at the screening visit, immediately after informed consent, up to the final visit/ETV



# TABLES OF CONTENTS

| | STATISTICAL ANALYSIS PLAN | 1 |
|---|---|---|
| | VERSIONS' HISTORY | 2 |
| | APPROVAL AND ACKNOWLEDGEMENT | 3 |
| | STUDY SCHEDULE | 5 |
| | TABLES OF CONTENTS | 7 |
| | ABBREVIATIONS | 9 |
| 1 | INTRODUCTION | 11 |
| 1.1 | Changes with respect to the study protocol | 11 |
| 2 | STUDY OBJECTIVES | 12 |
| 2.1 | Objectives | 12 |
| 2.1.1 | Primary objective | 12 |
| 2.1.2 | Secondary objectives | 12 |
| 2.2 | End-points | 12 |
| 2.2.1 | Primary end-point | 12 |
| 2.2.2 | Secondary end-points | 12 |
| 3 | INVESTIGATIONAL PLAN | 13 |
| 3.1 | Overall study design | 13 |
| 3.2 | Discussion of design | 13 |
| 4 | STUDY POPULATION | 14 |
| 4.1 | Target population | 14 |
| 4.2 | Inclusion criteria | 14 |
| 4.3 | Exclusion criteria | 14 |
| 4.3.1 | Not allowed treatments | 15 |
| 5 | STUDY SCHEDULE | 17 |
| 5.1 | Study visits and procedures | 17 |
| 5.2 | Diet and lifestyle | 20 |
| 5.3 | Restrictions | 21 |
| 5.4 | Protocol deviations | 21 |
| 6 | STUDY SUBJECT IDENTIFICATION METHOD AND TREATMENT ASSIGNMENT METHOD | 22 |
| 6.1 | Unique subject identifier | 22 |
| 6.2 | Subject identifier for the study | 22 |
| 6.3 | Randomisation | 22 |
| 6.4 | Treatment allocation | 22 |
| 6.5 | Blinding | 22 |
| 7 | STUDY EVALUATION PARAMETERS | 23 |
| 7.1 | Study variables | 23 |
| 7.1.1 | Primary variables | 23 |
| 7.1.2 | Secondary variables | 23 |
| 7.2 | PK assessments | 23 |
| 7.2.1 | PK parameters | 23 |
| 7.3 | Safety assessments | 24 |
| 7.4 | COVID-19 implications | 24 |
| 8 | STATISTICAL METHOD | 25 |
| 8.1 | Tables, listings and figures layout | 25 |





| 8.2 | Analysis sets | 25 |
|---|---|---|
| 8.2.1 | Definitions | 26 |
| 8.2.2 | Reasons for exclusion from the PK sets | 26 |
| 8.3 | Sample size and power considerations | 27 |
| 8.4 | Demographic, baseline and background characteristics | 27 |
| 8.4.1 | Subjects' disposition | 27 |
| 8.4.2 | <b>Analysis sets</b> | 27 |
| 8.4.3 | Subjects excluded from PK and/or safety analysis | 27 |
| 8.4.4 | Discontinued subjects | 27 |
| 8.4.5 | Protocol deviations | 27 |
| 8.4.6 | Treatment mismatch | 28 |
| 8.4.7 | Demography | 28 |
| 8.4.8 | Inclusion/exclusion criteria not met | 28 |
| 8.4.9 | Medical and surgical history | 28 |
| 8.4.10 | Prior and concomitant medication | 28 |
| 8.4.11 | Subjects' study visits | 28 |
| 8.4.12 | Fertility status and contraceptive method | 28 |
| 8.4.13 | Alcohol breath test, pregnancy test, SARS-COV2 test and urine drug test | 28 |
| 8.4.14 | Meals | 28 |
| 8.5 | IMP administration | 28 |
| 8.5.1 | IMP administration date/time | <b>2</b> 9 |
| 8.5.2 | Dose per body weight | <b>2</b> 9 |
| 8.5.3 | Wash-out | <b>2</b> 9 |
| 8.6 | PK analysis | <b>2</b> 9 |
| 8.6.1 | PK blood samples collection | <b>2</b> 9 |
| 8.6.2 | Descriptive pharmacokinetics | <b>2</b> 9 |
| 8.6.3 | Statistical comparison of pharmacokinetic parameters | 30 |
| 8.7 | Safety and tolerability analysis | 30 |
| 8.7.1 | Adverse events | 30 |
| 8.7.2 | Vital signs | 31 |
| 8.7.3 | Body weight | 31 |
| 8.7.4 | ECG | 31 |
| 8.7.5 | Laboratory data | 31 |
| 8.7.6 | Physical examination | 31 |
| 8.8 | Analysis datasets | 32 |
| 9 | REFERENCES | 33 |
| 10 | APPENDICES | 34 |



#### ABBREVIATIONS

β-HCG human chorionic gonadotropin β

 $\lambda_z$  Terminal elimination rate constant, calculated, if feasible, by log-linear regression

using at least 3 points

ADaM Analysis Data Model

AE Adverse Event

ANOVA Analysis of Variance

AUC<sub>0-t</sub> Area under the concentration-time curve from time zero to time t AUC $\infty$  Area under the concentration versus time curve up to infinity

%AUCextra Percentage of the residual area extrapolated to infinity in relation to the AUC∞

BLQL Below Lower Quantification Limit

BMI Body Mass Index BP Blood Pressure BT Body Temperature

CDISC Clinical Data Interchange Standards Consortium

CI Confidence Interval

C<sub>max</sub> Peak drug concentration

CPL Clinical Project Leader

CRA Clinical Research Associate

CRO Contract Research Organisation

CSR Clinical Study Report
CS Clinically Significant
CV Coefficient of Variation
DBP Diastolic Blood Pressure

ECG Electrocardiogram

eCRF electronic Case Report Form EMA European Medicines Agency ETV Early Termination Visit

FDA Food and Drug Administration

Frel Relative Bioavailability FSFV First Subject First Visit GCP Good Clinical Practice

HBs Ag Hepatitis B virus surface antigen HCV Ab Hepatitis C virus antibodies HIV Human Immunodeficiency Virus

HR Heart Rate

IB Investigator's Brochure

ICH International Conference on Harmonisation

IMP Investigational Medicinal Product INDs Investigational New Drug applications

IUD Intra-Uterine Device LSLV Last Subject Last Visit

MedDRA Medical Dictionary for Regulatory Activities

NC Not calculated

NDAs New Drug Applications

NSAIDs Non-Steroidal Anti-Inflammatory Drugs

OTC Over The Counter PE Point Estimate





PK Pharmacokinetics PT Preferred Term

PTAE Pre-Treatment Adverse Event

R Reference

SAP Statistical Analysis Plan SBP Systolic Blood Pressure SD Standard Deviation SOC System Organ Class

SOP Standard Operating Procedure SDTM Study Data Tabulation Model

SUSAR Suspected Unexpected Serious Adverse Reaction

T Test

TEAE Treatment-Emergent Adverse Event

THC delta-9-tetrahydrocannabinol

 $t_{1/2}$  Half-life

 $t_{max}$  Time to achieve  $C_{max}$ 

USDA United States Department of Agriculture

WHODDE World Health Organisation Drug Dictionary Enhanced




#### 1 INTRODUCTION

Statistical analysis will be performed by the Contract Research Organization (CRO) Biometry Unit. The end-points and methods of analysis specified in this SAP are consistent with ICH E6 (R2) and E9 guidelines (1, 2), with EMA guideline on the investigation of bioequivalence (3, 4) and on the investigation of drug interactions (5). The SAP has been compiled by the CRO Biometry Unit on the basis of the final version 1.0 of the clinical study protocol (6), reviewed by the Sponsor and finalized before the database lock.

# 1.1 Changes with respect to the study protocol

The following changes were introduced into the SAP with respect to the study protocol (6):

• the gender effect on bioavailability of ladarixin and its metabolites will be analysed for T and R separately using a non-parametric Wilcoxon signed ranks test on C<sub>max</sub>, AUC<sub>0-t</sub> and AUC<sub>0-∞</sub>. This analysis replaces the ANOVA including sequence, period, treatment, subject within sequence, sex and sex\*treatment interaction as fixed effect. The replacement has been done with the objective to better identify the gender effect when the same treatment is administered.



#### 2 STUDY OBJECTIVES

# 2.1 Objectives

#### 2.1.1 Primary objective

Primary objective of the study is to investigate the effect of food on the bioavailability of DF 2156Y after single dose administration of 400 mg of ladarixin to healthy male and female volunteers under fed and fasting conditions.

# 2.1.2 Secondary objectives

- to investigate the effect of gender on the bioavailability of DF 2156Y and its metabolites (DF 2108Y and DF 2227Y) after single dose administration of 400 mg of ladarixin to healthy male and female volunteers
- to evaluate safety and tolerability of a single dose administration of 400 mg ladarixin to healthy male and female volunteers

### 2.2 End-points

# 2.2.1 Primary end-point

• to evaluate and compare the rate (C<sub>max</sub>) and extent (AUC<sub>0-t</sub>; AUC<sub>0-∞</sub>) of absorption of DF 2156Y after single dose administration of 400 mg of ladarixin under fed and fasting conditions

# 2.2.2 Secondary end-points

- to evaluate and compare between genders the rate ( $C_{max}$ ) and extent ( $AUC_{0-t}$ ;  $AUC_{0-\infty}$ ) of absorption of DF 2156Y and its metabolites (DF 2108Y and DF 2227Y) after single dose administration of 400 mg of ladarixin to healthy male and female volunteers
- to describe the pharmacokinetic profile of DF 2156Y (total and unbound) and its metabolites (DF 2108Y and DF 2227Y) after single dose administration of 400 mg of ladarixin under fed and fasting conditions
- to collect safety and tolerability data of a single oral dose administration of 400 mg of ladarixin



#### 3 INVESTIGATIONAL PLAN

# 3.1 Overall study design

Single center, single dose, open label, randomized, two-way, crossover, food effect study.

# 3.2 Discussion of design

The study has been designed in agreement with the ICH E6 (R2) and E9 guidelines (1, 2), with EMA guideline on the investigation of bioequivalence (3, 4) and FDA guidance on the Assessing the Effects of Food on Drugs in INDs and NDAs (7).

The sample size was not calculated through any statistical calculation. The planned sample size is estimated as sufficient for the descriptive purposes of the study in compliance with the relevant EMA guideline for PK studies (3).

Each randomized subject will be allocated to a sequence of treatments (fasting [R] or fed [T]) in the two study periods (TR or RT) according to a computer generated randomization list.

The dose of 400 mg planned for the present study was selected because it proved to be well tolerated in the previous Phase I and II clinical studies (8).

The EMA Guideline on the Investigation of Drug Interactions (5) has been taken into account for the study administration of the IMP in fed conditions.

The wash-out interval of 14 days is considered appropriate according to the known half-life of ladarixin.

The open-label design was chosen since the study endpoints are based on the objective measurement of ladarixin and its active metabolites in plasma. The outcome variables are not influenced by the subjects or investigator being aware of the administered treatment.



#### 4 STUDY POPULATION

# 4.1 Target population

The study population included healthy volunteers (men and women), aged 18-55 years inclusive.

#### 4.2 Inclusion criteria

To be enrolled in this study, subjects had to fulfill all these criteria:

- 1. Informed consent: signed written informed consent before inclusion in the study
- 2. Sex and Age: men/women, 18-55 years old inclusive
- 3. Body Mass Index (BMI): 18.5-30 kg/m<sup>2</sup> inclusive
- 4. Vital signs: systolic blood pressure (SBP) 100-139 mmHg, diastolic blood pressure (DBP) 50-89 mmHg, heart rate (HR) 50-90 bpm and body temperature (BT) 35.5-37.5° C, measured after 5 min at rest in the sitting position
- 5. Full comprehension: ability to comprehend the full nature and purpose of the study, including possible risks and side effects; ability to co-operate with the investigator and to comply with the requirements of the entire study
- 6. Contraception and fertility (women only): women of child-bearing potential must not wish to get pregnant within 30 days after the end of the study and must be using at least one of the following reliable methods of contraception:
  - a. Hormonal oral, implantable, transdermal, or injectable contraceptives for at least 2 months before the screening visit until 30 days after final visit
  - b. A non-hormonal intrauterine device [IUD] or female condom with spermicide or contraceptive sponge with spermicide or diaphragm with spermicide or cervical cap with spermicide for at least 2 months before the screening visit until 30 days after final visit
  - c. A male sexual partner who agrees to use a male condom with spermicide until 30 days after final visit
  - d. A sterile sexual partner

Women participants of non-childbearing potential or in post-menopausal status for at least one year will be admitted.

For all women, pregnancy test result must be negative at screening and day -1.

#### 4.3 Exclusion criteria

Subjects meeting any of these criteria were not enrolled in the study:

- 1. Electrocardiogram (ECG) 12-leads (supine position): clinically significant abnormalities
- 2. *Physical findings*: clinically significant abnormal physical findings which could interfere with the objectives of the study



- 3. Laboratory analyses: clinically significant abnormal laboratory values indicative of physical illness
- 4. Allergy: ascertained or presumptive hypersensitivity to the active principles (ladarixin or derivatives) and/or formulations' ingredients; known hypersensitivity to non-steroidal anti-inflammatory drugs (NSAIDs); history of hypersensitivity to drugs (in particular methanesulfonyl propanamide) or allergic reactions in general, which the Investigator considers may affect the outcome of the study
- 5. *Diseases*: hypoalbuminemia or significant history of renal, hepatic, gastrointestinal, respiratory, skin, hematological, endocrine, neurological or cardiovascular diseases that may interfere with the aim of the study
- 6. *Medications*: medications, including over the counter drugs (in particular NSAIDs), herbal remedies and food supplements taken 14 days before the start of the study (in any case at least 5 times the half-life of the drug or a minimum of 14 days, whichever is longer), with the exception of paracetamol. Hormonal contraceptives and hormonal replacement therapy for women will be allowed
- 7. *Investigative drug studies:* participation in the evaluation of any investigational product for 3 months before this study. The 3-month interval is calculated as the time between the first calendar day of the month that follows the last visit of the previous study and the first day of the present study
- 8. Blood donation: blood donations for 3 months before this study
- 9. Drug, alcohol, caffeine, tobacco: history of drug, alcohol (>1 drink/day for women and >2 drinks/day for men, defined according to the USDA Dietary Guidelines 2015-2020], caffeine (>5 cups coffee/tea/day) or tobacco abuse (≥10 cigarettes/day)
- 10. SARS-COV2 test: positive SARS-COV2 test on day -3 or -2 of each study period
- 11. Positive to one of these test: Hepatitis B (HBs antigen), Hepatitis C (HCV antibodies), HIV 1/2 (HIV Ag/Ab combo) at screening.
- 12. Drug test: positive result at the drug test at screening or day -1 of each study period
- 13. Alcohol test: positive alcohol breath test at screening or day -1 of each study period
- 14. Diet: abnormal diets (<1600 or >3500 kcal/day) or substantial changes in eating habits in the 4 weeks before this study; vegetarians; vegans
- 15. Pregnancy (women only): positive or missing pregnancy test at screening or day -1 of each period, pregnant or lactating women

#### 4.3.1 Not allowed treatments

No medication, including over the counter drugs (in particular NSAIDs), herbal remedies and food supplements, is allowed for 14 days before the start of the study (in any case at least 5 times the half-life of the drug or a minimum of 14 days, whichever is longer), and during the whole study duration. Paracetamol is allowed as therapeutic counter-measure (maximum 2 g per day) for AEs according to the investigator's opinion. Hormonal contraceptives and hormonal replacement therapy for women are allowed.





The intake of any other medication is reported as a protocol deviation. However, it leads to subject's discontinuation from the study only if the investigator, together with the Sponsor, considers it could affect the study assessments or outcome.



#### 5 STUDY SCHEDULE

The schedule of the study is summarised at page 5.

## 5.1 Study visits and procedures

Each study subject undergoes 8 visits.

The study protocol foresees 2 periods separated by a wash-out interval of at least 14 days. Minimum study duration is 20 days, screening visit included. A written informed consent is obtained before any study assessment or procedure.

The first subject first visit (FSFV) is defined as the 1<sup>st</sup> visit performed at the Phase I Unit by the 1<sup>st</sup> screened subject. The last subject last visit (LSLV) is defined as the last visit performed at the Phase I Unit by the last subject, i.e. the last visit foreseen by the study protocol, independently of the fact that the subject is a completer or a withdrawn subject.

The following phases, visits and procedures are performed:

- Screening phase
  - Screening visit 1: between day -21 and day -2
  - Screening visit 1.1: day -3 or day -2
  - ➤ Period 1 visit 2: day -1
- Interventional phase
  - Period 1 visit 3: days 1-4
  - Wash-out interval of at least 14 days
  - Period 2 visit 4: day -3 or day -2
  - Period 2 visit 5: day -1
  - Period 2 visit 6: days 1-4
- Final phase
  - Final visit/early termination visit (ETV). In case of early discontinuation, discontinued subjects will undergo an ETV



| | Day | Procedures/Assessments | Notes |
|---|---|---|---|
| Screening – Visit 1 | From day -21<br>to day -2 | <ul> <li>Explanation to the subject of study aims, procedures and possible risks</li> <li>Informed consent signature</li> <li>Screening number (as S001, S002, etc.)</li> <li>Demographic data and life style recording</li> <li>Medical/surgical history</li> <li>Previous/concomitant medications</li> <li>Full physical examination (body weight, height, physical abnormalities)</li> <li>Vital signs measurement including blood pressure (BP), heart rate (HR) and body temperature (BT)</li> <li>ECG recording</li> <li>Laboratory analyses: hematology, blood chemistry, urinalysis, serum virology and serum pregnancy test (women only)</li> <li>Alcohol breath test</li> <li>Urine multi-drug kit test</li> <li>AE monitoring</li> <li>Inclusion/exclusion criteria evaluation</li> <li>Eligibility evaluation</li> </ul> | Note: The first two letters of the surname followed by the first two letters of the first name will be used in the Phase I Unit source document only and will not be transferred to the Sponsor. |
| Screening –<br>Visit 1.1 | Day -3 or -2 | <ul> <li>Nasal and pharyngeal swab for SARS-COV2 test</li> <li>Adverse events monitoring</li> <li>Previous/concomitant medications</li> </ul> | |
| Period 1 - Visit 2 | Day -1 | <ul> <li>Alcohol breath test</li> <li>Urine pregnancy test (women only)</li> <li>Urine multi-drug kit test</li> <li>ECG recording</li> <li>Vital signs measurement</li> <li>AE and concomitant medications</li> <li>Inclusion/exclusion criteria evaluation</li> <li>Eligibility evaluation</li> <li>Enrolment and randomization</li> </ul> | Arrival at the Phase I Unit in the evening. Confinement until the morning of day 4. Standardized low-fat dinner. Fasting for at least 10 h (overnight). |



| | Day | Procedures/Assessments | Notes |
|---|---|---|---|
| Period 1 - Visit 3 | Day I | <ul> <li>Investigational medicinal product administration at 8:00 ± 1 h</li> <li>Vital signs measurement at pre-dose</li> <li>ECG recording at pre-dose</li> <li>Blood sample collection for PK analysis at pre-dose (0) and 0.25 (15 min), 0.5 (30 min), 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12 and 18 h post-dose</li> <li>AE and concomitant medications</li> </ul> | Standardized high-fat and high caloric breakfast starting at 30 min predose for subjects receiving the investigational medicinal product under fed conditions in this study period. Breakfast must be completed within 30 min. Subjects receiving the investigational medicinal product under fasting conditions will not have breakfast. Standardized lunch and dinner at about 13:00 (5 h post-dose) and 20:00 (12 h post-dose), respectively |
| | Days 2 and 3 | <ul> <li>Blood sample collection for PK analysis at 24, 30, 36, 48, 54 and 60 h post-dose</li> <li>AE and concomitant medications</li> </ul> | Standardized breakfast, lunch and dinner at about 9:00, 13:00 and 20:00, respectively |
| | Day 4 | <ul> <li>Vital signs measurement upon discharge 72 h post-dose</li> <li>ECG recording upon discharge 72 h post-dose</li> <li>Blood sample collection for PK analysis at 72 h post-dose</li> <li>AE and concomitant medications</li> <li>Full physical examination (body weight and physical abnormalities) upon discharge</li> </ul> | Discharge from the Phase I Unit in the morning, after the 72-h post-dose blood sample collection, ECG recording, vital signs check and full physical examination. Upon leaving, the subjects will be instructed to contact immediately the investigator in case of occurrence of any adverse reactions. |
| Wash-out | At least 14<br>days | A wash-out interval of at least 14 days between the two administrations of the two study periods | |
| Period 2 - Visit 4 | Day -3 or -2 | As visit 1.1, day -3 or -2 | |



| | Day Procedures/Assessments | | Notes |
|---|---|---|---|
| Period 2 - Visit 5 | Day -1 | As visit 2, excluding enrolment and randomization. In addition full physical examination (body weight and physical abnormalities) will be performed. | As visit 2 |
| Period 2 - Visit 6 | Days 1-4 | As visit 3. IMP administered according to the randomization list and crossover design | As visit 3 |
| Final Visit/ETV | Day 4 of<br>period 2<br>/at ETV in case<br>of<br>discontinuation | <ul> <li>Full physical examination (body weight and physical abnormalities; also vital signs and ECG in case of ETV)</li> <li>Alcohol breath test</li> <li>Urine multi-drug kit test</li> <li>Laboratory analyses as at screening, with the exception of virology, coagulation, microbiology, albumin and globulin</li> <li>AEs and concomitant medications</li> <li>In case of clinically significant results at the final visit, the subjects will be followed-up by the investigator until the normalization of the concerned clinical parameter(s)</li> </ul> | Upon leaving, the subjects will be instructed to contact immediately the investigator in case of occurrence of any adverse reactions. |

#### 5.2 Diet and lifestyle

On day -1 of each period, a standardized low-fat dinner is served after confinement. On day 1 of each study period, all the subjects do not take any food or drinks (except water) for at least 10 h (i.e. overnight). The subjects allocated to the fed conditions, after the overnight fasting period, receive a high-fat and high-caloric breakfast [see § 6.2.1 of the study protocol (6) for details] starting 30 min pre-dose and complete their breakfast within 30 min, while the subjects allocated to the fasting conditions fast overnight and then receive their treatment. Water is allowed as desired, except for 1 h before and 1 h after IMP administration. In order to maintain an adequate hydration, the subjects are encouraged to drink at least 150 mL of still mineral water every 2 h for 5 h post-dose, starting at 1 h post-dose.

On day 1, all subjects remain fasted until 5 h post-dose. A standardized lunch and dinner is served at approximately 5 h and 12 h post-dose (at approximately 13:00 and 20:00). On days 2 and 3, standardized breakfast, lunch and dinner are served to all subjects at about 9:00, 13:00 and 20:00, respectively.

One cup of coffee or tea is allowed after each meal only; any other coffee, tea or food containing xanthines (i.e. coke, chocolate, etc.), alcohol and grapefruit is forbidden during confinement. In particular, grapefruit and alcohol are forbidden for 24 h before the first IMP administration until the end of the study.





The subjects are allowed to smoke 9 cigarettes during confinement, one after each meal, with the exclusion of the high-fat and high-caloric breakfast.

During confinement, routine ambulant daily activities are strongly recommended.

#### 5.3 Restrictions

During each study period, the subjects are confined from the evening preceding the IMP administration (study day -1) until the morning of day 4.

For the 4 h following the administration, when not involved in study activities, the subjects remain seated. They are not allowed to lie down.

During confinement, hazardous, strenuous or athletic activities are not permitted.

#### 5.4 Protocol deviations

All un-intended departures from the approved protocol, from other agreed study documents, from relevant ICH guidelines, from other applicable regulatory requirements or from SOPs will be treated as deviations.

A deviation is defined major when it is significant and could, indirectly or over time, negatively influence the quality or the authenticity of the data, or the privacy, safety and security of the participants in a clinical trial.



# 6 STUDY SUBJECT IDENTIFICATION METHOD AND TREATMENT ASSIGNMENT METHOD

# 6.1 Unique subject identifier

All the subjects who sign the informed consent form for the present study are coded with "unique subject identifiers" when data are extracted from the study database into the domains of the CDISC SDTM model. The unique subject identifier consists of the sponsor study code (i.e. LDX0219), the 3-digit site number (i.e. 001), the 4-digit screening number (e.g. S001, S002, etc.) and, if applicable, the 3-digit subject randomization number (e.g. 001, 002, etc.). Study code, site number, screening number and subject randomization number are separated by slashes ("/") [example: LDX0219/001/S001/001].

# 6.2 Subject identifier for the study

The last 8 digits of the unique subject identifier (enrolled subjects), corresponding to the subject screening and subject randomization numbers separated by a slash, or the last 4 digits of the unique subject identifier (not enrolled subjects), corresponding to the subject screening number, will appear as subject identifier in the individual listings and figures of the CSR and will be used to identify the subjects in in-text tables or wording (if applicable).

#### 6.3 Randomisation

The randomization list was computer-generated by the Biometry Unit of the CRO, using the PLAN procedure of SAS® version 9.3 (TS1M1) (9). The randomization list was supplied to the study site before study start and will be attached to the final CSR.

Randomization was stratified by sex in order to have the same number of men and women for every sequence of treatments.

#### 6.4 Treatment allocation

Subjects were assigned to one sequence of treatments (e.g. TR or RT) i.e. to receive the IMP in fed conditions (T treatment) during period 1 and in fasting conditions (R treatment) in period 2 or vice versa according to their randomization number.

Randomization number was given to the subjects on study Day -1 of period 1 and was used to assign the treatment sequence.

## 6.5 Blinding

This is an open-label trial. No masking procedure will be applied since an open-label design was considered adequate for evaluating objective measures such as pharmacokinetic parameters. All the personnel involved in the analytical determinations of ladarixin and its metabolites in plasma samples collected from the volunteers will be maintained in blind conditions.



#### 7 STUDY EVALUATION PARAMETERS

# 7.1 Study variables

#### 7.1.1 Primary variables

 $C_{max}$  and  $AUC_{0-t}$  of plasma DF 2156Y after single dose administration of 400 mg of ladarixin under fed and fasting conditions.

#### 7.1.2 Secondary variables

- AUC<sub>0- $\infty$ </sub>,  $t_{max}$ ,  $t_{1/2}$ ,  $\lambda_z$  and  $F_{rel}$  of plasma DF 2156Y after single dose administration of 400 mg of ladarixin under fed and fasting conditions
- $C_{max}$ ,  $AUC_{0-t}$ ,  $AUC_{0-\infty}$ ,  $t_{max}$ ,  $t_{1/2}$ ,  $\lambda_z$  and  $F_{rel}$  of plasma DF 2156Y and its metabolites (DF 2108Y and DF 2227Y) after single dose of 400 mg of ladarixin under fed and fasting conditions measured and calculated in healthy men and healthy women
- Treatment-emergent adverse events (TEAEs), vital signs (BP, HR, BT), body weight, ECGs, physical examinations, laboratory parameters (hematology, blood chemistry and urine analysis)

#### 7.2 PK assessments

The following PK parameters will be measured and/or calculated for DF 2156Y and its metabolites, DF 2108Y and DF 2227Y.

#### 7.2.1 PK parameters

C<sub>max</sub>: Maximum plasma concentration

 $t_{max}$ : Time to achieve  $C_{max}$ 

 $\lambda_z$ : Terminal rate constant, calculated, if feasible, by log-linear regression using at

least 3 points

 $t_{1/2}$ : Half-life, calculated, if feasible, as  $\ln 2/\lambda_z$ 

 $AUC_{0-t}$ : Area under the concentration-time curve from administration to the last

observed concentration time t, calculated with the linear trapezoidal method

 $AUC_{0-\infty}$ : Area under the concentration-time curve extrapolated to infinity, calculated, if

feasible, as  $AUC_{0-t} + C_t/\lambda_z$ , where  $C_t$  is the last measurable drug concentration

%AUC<sub>extra</sub>: Percentage of the residual area  $(C_t/\lambda_z)$  extrapolated to infinity in relation to the

total AUC<sub>0- $\infty$ </sub>, calculated, if feasible, as  $100 \times [(C_t/\lambda_z)/AUC_{0-\infty}]$ 

 $F_{rel}$ : Relative bioavailability, calculated as ratio  $AUC_{0-t}(T)/AUC_{0-t}(R)$ 



The sampling schedule is considered adequate if the ratio  $AUC_{0-t}/AUC_{0-\infty}$  equals or exceeds a factor of 0.8 (i.e. if % $AUC_{extra}$  is <20%) for more than 80% of the individual PK profiles. This assures that the primary variable  $AUC_{0-t}$  covers a sufficient percentage of the theoretical total extent of exposure. AUC truncated at 72 h ( $AUC_{0-72h}$ ) may be used as an alternative to  $AUC_{0-t}$  for comparison of extent of exposure as the absorption phase has been covered by 72 h for immediate release formulations.

The quality of log-linear regression (and, consequently, the reliability of the extrapolated PK parameters) should be demonstrated by a determination coefficient  $R^2 > 0.8$ . Individual extrapolated parameters, when considered unreliable, will be reported as NC (not calculated).

# 7.3 Safety assessments

Safety and general tolerability of the IMP will be based on TEAEs, physical examinations including body weight, vital signs, routine hematology, blood chemistry, urinalysis laboratory tests and ECGs.

# 7.4 COVID-19 implications

The presence of protocol deviations and/or adverse events related to the COVID-19 pandemic will be captured and listed in the same listings, but with a clear description identifying the COVID-19 pandemic relationship.



#### 8 STATISTICAL METHOD

The statistical analysis of demographic, baseline and background characteristics, safety and tolerability data will be performed using SAS® version 9.3 (TS1M1) (9).

The PK analysis and the statistical analysis of PK parameters will be performed using Phoenix WinNonlin<sup>®</sup> version 6.3 (10) and SAS<sup>®</sup> version 9.3 (TS1M1).

The data documented in this study and the parameters measured will be evaluated and compared using classic descriptive statistics, i.e. geometric mean (PK data only), arithmetic mean, SD, CV (%), minimum, median and maximum values for quantitative variables and frequencies for qualitative variables.

Not available data will be evaluated as "missing values".

## 8.1 Tables, listings and figures layout

Tables, listings and figures will be provided according to the following settings:

Background: WhiteForeground: BlackFont face: TimesFont style: Roman

• Font size: 10 pt

• Font weight: Medium (data, footers and notes), Bold (titles and headers)

Font width: Normal
Layout: Landscape
Top Margin: 2.5 cm
Bottom Margin: 2.5 cm

Left Margin: 0.8 cmRight Margin: 0.8 cm

• Test label: Ladarixin fed (T)

• Reference label: Ladarixin fasting (R)

• Date format: ddMMMyyyy

- Means, standard deviations, percent coefficient of variations, medians, lower confidence limits and upper confidence limits will be rounded to one digit more than the original data
- Minima and maxima will keep the same number of decimal digits as the source values
- Two-sided p-values will be rounded to the fourth decimal digit and will be flagged by an asterisk (\*) in case of statistical significance (i.e. p-value < 0.05 or, in case of centre by treatment interaction, p-value < 0.10)
- p-values lower than 0.0001 will be reported as "<.0001 \*".

The data and results of Ladarixin fed (T) will be presented before the data and results of Ladarixin fasting (R) in all listings and tables.

# 8.2 Analysis sets



#### 8.2.1 Definitions

A subject will be defined as <u>screened</u> after the signature of the informed consent, regardless of the completion of all the screening procedures.

A subject will be defined as eligible if he/she meets all the inclusion/exclusion criteria. Otherwise he/she will be defined as a screen failure.

A subject will be defined as <u>enrolled</u> in the study if he/she is included into the interventional phase of the study. The enrolment will be performed through randomised allocation to one treatment sequence.

An eligible but not enrolled subject will be defined as a <u>reserve</u>.

In the present study, randomized subjects will be the same as enrolled subjects.

Analysis sets are defined as follows:

- Enrolled set: all enrolled subjects. This analysis set will be used for demographic, baseline and background characteristics
- Safety set: all subjects who receive at least one dose of study treatments. This analysis set will be used for the safety and tolerability analyses
- PK set 1: all subjects randomized who fulfill the study protocol requirements in terms of investigational treatment intake and have evaluable PK data readouts for DF 2156Y with no major deviations that may affect the PK results. This analysis set will be used for the statistical analysis of the PK results for DF 2156Y.
- PK set 2: all subjects randomized who fulfill the study protocol requirements in terms of investigational treatment intake and have evaluable PK data readouts for DF 2108Y and DF 2227Y, with no major deviations that may affect the PK results. This analysis set will be used for the statistical analysis of the PK results for DF 2108Y and DF 2227Y.

Each subject will be coded by the CRO Biometry Unit as valid or not valid for the safety set and the PK sets. Subjects will be evaluated according to the treatment they actually receive.

# **8.2.2** Reasons for exclusion from the PK sets

Reasons for the exclusion of subjects from the PK sets before the bioanalysis are the following:

- vomiting and diarrhea before or after drug intake which could render the plasma concentration-time profile unreliable
- intake of concomitant medications which could render the plasma concentration-time profile unreliable
- AEs which could render the plasma concentration-time profile unreliable
- administration errors which could render the plasma concentration-time profile unreliable
- other events which could render the plasma concentration-time profile unreliable If one of these events occurred, it was to be noted in the eCRF as the study was being conducted.



Reason for the exclusion of subjects from the PK sets after the bioanalysis is the following:

• in case of more than 5 randomized patients affected by COVID-19 during the study, these subjects will be excluded from the Statistical comparison of PK parameters (§8.6.3)

# 8.3 Sample size and power considerations

The sample size was not calculated through any statistical calculation. A sample size of 36 subjects (18 men and 18 women) was estimated as sufficient for the descriptive purposes of the present study in compliance with the relevant EMA guideline for PK studies (3).

Drop-out subjects will not be replaced.

## 8.4 Demographic, baseline and background characteristics

Demographic, baseline and background characteristics will be reported for all the enrolled subjects and analyses will be performed according to the treatment they actually received.

### 8.4.1 Subjects' disposition

The disposition of all subjects enrolled in the study will be listed (Listing 16.2.4.1) and summarised (Table 14.1.1.1). The number and proportion of subjects enrolled, treated and completing the study, the number and proportion of withdrawals and the reasons for withdrawal will be presented.

#### 8.4.2 Analysis sets

The subjects included in each analysis sets will be listed (Listing 16.2.4.2) and summarised by treatment group (Table 14.1.1.2).

#### 8.4.3 Subjects excluded from PK and/or safety analysis

All subjects excluded from the PK and/or safety analysis will be listed (Listing 16.2.3.1) and the reasons for exclusion will be reported.

#### 8.4.4 Discontinued subjects

All subjects who discontinued the clinical trial (if any) will be listed (Listing 16.2.1.1). Last IMP administered before discontinuation, gender, age, last visit performed before discontinuation, time elapsed from last IMP administration (days), date of premature discontinuation and primary reason for subject premature discontinuation will be reported.

#### 8.4.5 Protocol deviations

All the protocol deviations reported during the clinical trial will be listed (Listing 16.2.2.1) and summarised by severity (major and minor) (Table 14.1.1.5). The number and proportion of subjects for each deviation will be reported.



#### 8.4.6 Treatment mismatch

All subjects with actual treatment sequence different from the assigned one will be listed (Listing 16.2.2.2).

# 8.4.7 **Demography**

Demographic data will be listed (Listing 16.2.4.3) and summarised (Table 14.1.1.3). The number and proportion of subjects in each category for categorical variables (e.g. gender, race) and descriptive statistics (mean, SD, CV%, minimum, median and maximum) for continuous variables (e.g. age, weight) will be presented.

#### 8.4.8 Inclusion/exclusion criteria not met

All the unmet inclusion/exclusion criteria will be listed (Listing 16.2.4.4) and summarised (Table 14.1.1.4).

## 8.4.9 Medical and surgical history

All the diseases of medical history and the surgeries of all subjects enrolled in the study will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) version 23.1 and listed (Listing 16.2.10.1).

#### 8.4.10 Prior and concomitant medication

All prior and concomitant medications will be coded using the World Health Organization Drug Dictionary Enhanced (WHODDE) version March 2020 and listed (Listing 16.2.10.3).

#### 8.4.11 Subjects' study visits

The dates of all subjects study visits will be listed (Listing 16.2.10.4).

#### 8.4.12 Fertility status and contraceptive method

The fertility status and the contraceptive method used by the subjects will be listed (Listing 16.2.10.5).

#### 8.4.13 Alcohol breath test, pregnancy test, SARS-COV2 test and urine drug test

The date/time and the result of alcohol breath test, pregnancy test, SARS-COV2 test and urine drug test will be listed (Listing 16.2.8.1).

#### **8.4.14** Meals

The start date/time of the standardised meals will be listed (Listing 16.2.10.6).

#### 8.5 IMP administration



#### 8.5.1 IMP administration date/time

The date and time of all IMP administrations will be listed (Listing 16.2.5.1).

# 8.5.2 Dose per body weight

The dose per body weight of ladarixin will be listed (Listing 16.2.5.2) and summarised using descriptive statistics (Table 14.3.5.6).

The body weight collected at the screening visit will be used for the calculation.

#### 8.5.3 Wash-out

The minimum and maximum number of days of wash-out between periods will be presented (Table 14.3.5.7).

# 8.6 PK analysis

The PK analysis will be performed on the subjects included into the PK Sets.

Subjects will be analysed according to the treatment they actually received.

# 8.6.1 PK blood samples collection

The actual date/time of PK blood samples collection will be listed (Listing 16.2.5.3).

# 8.6.2 Descriptive pharmacokinetics

A descriptive PK will be presented for plasma total and unbound DF 2156Y and its metabolites DF 2108Y and DF 2227Y.

Individual subject concentrations of total and unbound DF 2156Y and its metabolites DF 108Y and DF 2227Y will be presented in data listings (Listing 16.2.5.4, Listing 16.2.5.5, Listing 16.2.5.6, Listing 16.2.5.7) and summarised at each time point by treatment (Table 14.2.1.1, Table 14.2.1.2, Table 14.2.1.3, Table 14.2.1.4).

Individual (figures in section 16.2.5) and mean curves (+SD at sampling times) (figures in section 14.2.1), indicating inter-subject variability, will be plotted. Mean curves will be presented by treatment and by treatment and sex.

PK parameters of total plasma DF 2156Y and its metabolites DF 2108Y and DF 2227Y will be listed (Listing 16.2.6.1, Listing 16.2.6.2, Listing 16.2.6.3, Listing 16.2.6.4) and summarised by treatment and by treatment and sex (Table 14.2.2.1, Table 14.2.2.2, 14.2.2.3, 14.2.2.4).

Data below the lower quantification limit (BLQL) will be considered as 0 in the calculations and presented as BLQL in listings and tables. As a consequence of BLQL (i.e. 0) values, calculated geometric means (if requested) could be null. For this reason, in the presence of any null value, the geometric mean will be reported as NC. If for an individual PK curve, a log-linear regression with a correlation coefficient  $R^2 > 0.8$  cannot be obtained, the



extrapolated PK parameters will be reported as NC and considered missing in the calculations of descriptive statistics.

#### 8.6.3 Statistical comparison of pharmacokinetic parameters

For the primary end-point evaluation of food effect,  $C_{max}$ ,  $AUC_{0-t}$  and  $AUC_{0-\infty}$  of total plasma DF 2156Y will be compared between fed and fasting conditions (T vs. R) using analysis of variance (ANOVA) for a cross-over design on log-transformed data for evaluation of the food effect. Period, treatment, sequence and subject within sequence will be taken in account as sources of variation and they will be treated as fixed effect (Table 14.2.3.1).

The 90% confidence intervals (CI) will be calculated for the point estimates (PE, i.e. the T/R ratio of least square geometric means) of the PK parameters.

Established criteria for the absence of a food effect are that the 90% CI for the T/R ratio of the geometric means of the PK parameters under consideration are within the 80.00-125.00% range.

For the purpose of exploring the gender effect on bioavailability of ladarixin and its metabolites,  $C_{max}$ ,  $AUC_{0-t}$  and  $AUC_{0-\infty}$  of total plasma DF 2156Y and of DF 2108Y and DF 2227Y will be analysed for T and R separately using a non-parametric Wilcoxon signed ranks test (Table 14.2.3.2, Table 14.2.3.3, Table 14.2.3.4).

### 8.7 Safety and tolerability analysis

The safety and tolerability analysis will be performed on the subjects included into the Safety Set.

Subjects will be analysed according to the treatment they actually received.

# 8.7.1 Adverse events

AEs will be coded by System Organ Class (SOC) and Preferred Term (PT), using the Medical Dictionary for Regulatory Activities (MedDRA).

AEs will be classified as pre-treatment AEs (PTAEs) and TEAEs, according to the period of occurrence, as follows:

- PTAEs: all AEs occurring after informed consent signature by the enrolled subject but before the first dose of IMP and not negatively affected by the first dose of IMP
- TEAEs: all AEs occurring or worsening after the administration of the first dose of IMP

Individual PTAEs and TEAEs will be listed in subject data listings (Listing 16.2.7.2, Listing 16.2.7.1). No summary table will be provided for PTAEs.

TEAEs will be summarised by treatment group and overall. The number and percentage of subjects with any TEAE and the number of TEAEs will be tabulated by SOC and PT, seriousness, relationship to treatment and severity.



For TEAEs that change intensity during the study (e.g. from mild to moderate or from moderate to mild), the most severe intensity will be reported in the summary tables (Table 14.3.1.1, Table 14.3.1.2, Table 14.3.1.3, Table 14.3.1.4).

Should any serious TEAE occur, the number and percentage of subjects with any serious TEAE, the number of serious TEAEs, the number and percentage of subjects with any serious TEAE related to study drug and the number of serious TEAEs related to study drug will be presented (Table 14.3.1.5, Table 14.3.1.6).

All TEAEs leading to death will be listed, all Serious TEAEs will be listed and all TEAEs leading to discontinuation will be listed, if applicable (Table 14.3.2.1).

# 8.7.2 Vital signs

The date/time of vital signs assessments and the values of vital signs will be listed (Listing 16.2.9.1) and summarised using descriptive statistics at screening, day -1 and end of study (Table 14.3.5.2) and by treatment during the study (Table 14.3.5.3).

A table of all the abnormal vital signs' values will be presented (Table 14.3.5.1).

## 8.7.3 Body weight

Body weight values will be listed (Listing 16.2.9.1) and summarised using descriptive statistics at screening and end of study (Table 14.3.5.2).

#### 8.7.4 ECG

The date/time of ECG assessments and the overall investigator's interpretation (as normal, abnormal, not clinically significant or abnormal, clinically significant) and all abnormalities found (if any) will be listed (Listing 16.2.9.2, Listing 16.2.9.3).

The overall investigator's interpretations will be summarised using contingency tables at screening, day -1 and end of study (Table 14.3.5.4) and by treatment during the study (Table 14.3.5.5).

#### 8.7.5 Laboratory data

Date/time of samples collection, overall Investigator's interpretation (as normal or abnormal and, if abnormal, clinically significant or not clinically significant) and clinically significant findings (if any) will be listed (Listing 16.2.8.2).

All laboratory results will be listed (Listing 16.2.8.1) and a table of all the abnormal values will be presented (Table 14.3.4.1). The overall Investigator's interpretation will be summarised using tables of frequency (Table 14.3.4.2).

#### 8.7.6 Physical examination

Date of the physical examination, overall Investigator's interpretation (as normal or abnormal and, if abnormal, clinically significant or not clinically significant) and clinically significant abnormalities (if any) will be listed (Listing 16.2.10.2).





# 8.8 Analysis datasets

Analysis datasets will be created according to the version 2.1 of the ADaM model of CDISC (11).



#### 9 REFERENCES

- 1 ICH Topic E6 (R2): Good clinical practice.
- 2 ICH Topic E9: Statistical principles for clinical trials.
- Guidance on the investigation of bioequivalence. CPMP/EWP/QWP/1401/98 Rev. 1/Corr \*\*, 20 January 2010
- 4 Questions & Answers: Positions on specific questions addressed to the pharmacokinetics working party. EMA/618604/2008 Rev. 8, 10 October 2013
- 5 Guideline on the investigation of drug interactions. CPMP/EWP/560/95/Rev. 1 Corr. 2\*\*, 21JUN2012
- 6 Study Protocol CRO-PK-20-345. "Influence of Food on the Oral Bioavailability of Ladarixin 200 mg Capsule in Healthy Volunteers of Both Sexes. A Single dose (400 mg), Randomized, Open Label, Two-Way Crossover Study". Final version 1.0, 28MAY2020
- Guidance for industry. Assessing the Effects of Food on Drugs in INDs and NDAs—Clinical Pharmacology Considerations. U.S. Department of Health and Human Services, Food and Drug Administration, Center for Drug Evaluation and Research. CDER, February 2019
- 8 Dompé, Ladarixin (DF 2156A formerly meraxin) Investigator's Brochure, final version No. 7, 09APR20
- 9 SAS/STAT® User's Guide
- 10 Phoenix 1.3 User's Guide, Pharsight Corporation
- 11 CDISC Analysis Data Model Version 2.1





# 10 APPENDICES

- 1. Section 14 Tables Shells
- 2. Section 16.2 Individual Subject Data Listings Shells



#### Section 14 - Tables Shells

| Table 14.1.1.1 | - Subjects' | disposition - | Enrolled set |
|----------------|-------------|---------------|--------------|

- Table 14.1.1.2 Analysis sets Enrolled set
- Table 14.1.1.3 Demography Enrolled set, Safety set, PK set 1 and PK set 2
- Table 14.1.1.4 Inclusion/exclusion criteria not met Enrolled set, Safety set, PK set 1 and PK set 2
- Table 14.1.1.5 Protocol deviations Enrolled set, Safety set, PK set 1 and PK set 2
- Table 14.2.1.1 Total DF 2156Y concentrations (µg/mL) measured in plasma PK Set 1
- Table 14.2.1.2 Unbound DF 2156Y concentrations (µg/mL) measured in plasma PK Set 1
- Table 14.2.1.3 DF 2108Y concentrations (µg/mL) measured in plasma PK Set 2
- Table 14.2.1.4 DF 2227Y concentrations (µg/mL) measured in plasma PK Set 2
- Table 14.2.2.1 Total DF 2156Y plasma PK parameters PK Set 1
- Table 14.2.2.2 DF 2108Y plasma PK parameters PK Set 2
- Table 14.2.2.3 DF 2227Y plasma PK parameters PK Set 2
- Table 14.2.2.4 Total DF 2156Y, DF 2108Y and DF 2227Y relative bioavailability in plasma calculated as AUC0-t T/R ratio PK Sets 1 and 2
- Table 14.2.3.1 Statistical analysis on total DF 2156Y plasma PK parameters PK set 1
- Table 14.2.3.2 Statistical analysis of gender effect on total DF 2156Y plasma PK parameters PK set 1
- Table 14.2.3.3 Statistical analysis of gender effect on DF 2108Y plasma PK parameters PK set 2
- Table 14.2.3.4 Statistical analysis of gender effect on DF 2227Y plasma PK parameters PK set 2
- Table 14.3.1.1 Global incidence of subjects with treatment-emergent adverse events Safety set
- Table 14.3.1.2 Subjects with treatment-emergent adverse events by system organ class and preferred term Safety set
- Table 14.3.1.3 Subjects with treatment-emergent adverse events by intensity, system organ class and preferred term Safety set
- Table 14.3.1.4 Subjects with treatment-emergent adverse events related to the IMP by system organ class and preferred term Safety set
- Table 14.3.1.5 Subjects with serious treatment-emergent adverse events by system organ class and preferred term Safety set
- Table 14.3.1.6 Subjects with serious treatment-emergent adverse events related to the IMP by system organ class and preferred term Safety set
- Table 14.3.2.1 Treatment emergent adverse events leading to death, serious adverse events or treatment emergent adverse events leading to discontinuation Safety set
- $Table\ 14.3.4.1 \text{ -} Abnormal\ laboratory\ values \text{ -} Safety\ set}$
- Table 14.3.4.2 Contingency tables of investigator's interpretation of laboratory test results Safety set
- Table 14.3.5.1 Abnormal vital signs Safety set
- Table 14.3.5.2 Descriptive statistics of vital signs and body weight at screening, day -1 and end of study Safety set
- Table 14.3.5.3 Descriptive statistics of vital signs during the study Safety set
- Table 14.3.5.4 Contingency tables of investigator's interpretation of ECG at screening, day -1 and end of study Safety set

CROSS Research S.A.

Statistical analysis plan CRO-PK-20-345

Sponsor code LDX0219
Ladarixin 200 mg capsules - food effect
Final version 1.0, 10FEB21



Section 14 - Tables Shells

Table 14.3.5.5 - Contingency tables of investigator's interpretation of ECG during the study - Safety set

Table 14.3.5.6 - Descriptive statistics of dose per body weight - Safety set

Table 14.3.5.7 - Descriptive statistics of wash-out - Safety set



### Table 14.1.1.1 - Subjects' disposition - Enrolled set

| | Overall<br>n (%) |
|--------------------------------------------|------------------|
| Enrolled | nn (xx.x) |
| Discontinued before treatment <sup>1</sup> | nn(xx.x) |
| Treated <sup>1</sup> | nn(xx.x) |
| Completed <sup>2</sup> | nn(xx.x) |
| Discontinued <sup>2</sup> | nn(xx.x) |
| Adverse event <sup>2</sup> | nn(xx.x) |
| Withdrawal by subject <sup>2</sup> | nn(xx.x) |

Note: The number and the proportion of subjects of each disposition event are reported Note 1: The denominator for calculating the proportions is the number of enrolled subjects

Note 2: The denominator for calculating the proportions is the number of enrolled and treated subjects

Source: Listing 16.2.4.1 - Subjects' disposition

Program: Tables\k345-ds-tbl.sas



### Table 14.1.1.2 - Analysis sets - Enrolled set

| | | <b>Enrolled Set</b> | |
|---|---|---|---|
| | Ladarixin<br>fed (T)<br>N=XX<br>n (%) | Ladarixin<br>fasting (R)<br>N=XX<br>n (%) | Overall<br>N=XX<br>n (%) |
| Safety Set | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| PK Set 1 | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| PK Set 2 | nn (xx.x) | nn (xx.x) | nn (xx.x) |

Note: Subjects are summarised according to the product they were assigned to

The number and the proportion of subjects included in each analysis set are reported

The denominator for calculating the proportions is the number of subjects in the enrolled set of each treatment group and overall

Source: Listing 16.2.4.2 - Analysis sets

 $Program: Tables \backslash k345\text{-}ds\text{-}tbl.sas$ 



Table 14.1.1.3 - Demography - Enrolled set, Safety set, PK set 1 and PK set 2

| | | Statistics | Enrolled Set<br>N=XX | Safety Set<br>N=XX | PK Set 1<br>N=XX | PK Set 2<br>N=XX |
|---|---|---|---|---|---|---|
| Sex | Female | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Male | n (%) | nn(xx.x) | nn (xx.x) | nn (xx.x) | nn(xx.x) |
| Race | American Indian or Alaska Native | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Asian | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Native Hawaiian or Other Pacific Islander | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Black or African American | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | White | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Other | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Age (years) | | N | nn | nn | nn | nn |
| | | Mean | XX.X | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X | XX.X |
| | | CV% | XX.X | XX.X | XX.X | XX.X |
| | | Min | XX | XX | XX | XX |
| | | Median | XX.X | XX.X | XX.X | XX.X |
| | | Max | XX | XX | XX | XX |
| Weight (kg) | | N | nn | nn | nn | nn |
| 2 ( 3) | | Mean | XX.XX | XX.XX | XX.XX | XX.XX |
| | | SD | XX.XX | XX.XX | XX.XX | XX.XX |
| | | CV% | XX.XX | XX.XX | XX.XX | XX.XX |
| | | Min | XX.X | XX.X | XX.X | XX.X |
| | | Median | XX.XX | XX.XX | XX.XX | XX.XX |
| | | Max | XX.X | XX.X | XX.X | XX.X |

Note: The number and the proportion of subjects of each sex and race are reported

The denominator for calculating the proportions is the number of subjects in each analysis set

Source: Listing 16.2.4.3 - Demography

 $Program: Tables \verb|\k345-dm-tbl.sas|$ 



Table 14.1.1.3 - Demography - Enrolled set, Safety set, PK set 1 and PK set 2

| | Statistics | Enrolled Set<br>N=XX | Safety Set<br>N=XX | PK Set 1<br>N=XX | PK Set 2<br>N=XX |
|---|---|---|---|---|---|
| Body Mass Index (kg/m²) | N | nn | nn | nn | nn |
| | Mean | XX.XX | XX.XX | XX.XX | XX.XX |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX |
| | CV% | XX.XX | XX.XX | XX.XX | XX.XX |
| | Min | XX.X | XX.X | XX.X | XX.X |
| | Median | XX.XX | XX.XX | XX.XX | XX.XX |
| | Max | XX.X | XX.X | XX.X | XX.X |

Note: The number and the proportion of subjects of each sex and race are reported

The denominator for calculating the proportions is the number of subjects in each analysis set

Source: Listing 16.2.4.3 - Demography Program: Tables\k345-dm-tbl.sas



Table 14.1.1.4 - Inclusion/exclusion criteria not met - Enrolled set, Safety set, PK set 1 and PK set 2

| | Enrolled Set | Safety Set | PK Set 1 | PK Set 2 |
|---|---|---|---|---|
| | N=XX | N=XX | N=XX | N=XX |
| Number of subjects with any inclusion/exclusion criteria not met | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Inclusion | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Inclusion criterion 1 Inclusion criterion 2 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Exclusion | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Exclusion criterion 1 Exclusion criterion 2 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |

Note: The number and the proportion of subjects for any criterion not met are reported

The denominator for calculating the proportions is the number of subjects in each analysis set

Source: Listing 16.2.4.4 - Inclusion/Exclusion criteria not met

 $Program: Tables \verb|\k345-ie-tbl.sas|$ 



Table 14.1.1.5 - Protocol deviations - Enrolled set, Safety set, PK set 1 and PK set 2

| | Enrolled Set<br>N=XX | Safety Set<br>N=XX | PK Set 1<br>N=XX | PK Set 2<br>N=XX |
|---|---|---|---|---|
| Number of subjects with any protocol deviation | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Major | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Treatment deviation | nn(xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Inclusion criteria violation | nn(xx.x) | nn (xx.x) | nn(xx.x) | nn(xx.x) |
| Exclusion criteria violation | nn(xx.x) | nn (xx.x) | nn(xx.x) | nn(xx.x) |
| Medication not admitted | nn(xx.x) | nn(xx.x) | nn (xx.x) | nn(xx.x) |
| Minor | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Deviation from scheduled sampling time | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | <del></del> | ••• | ••• | ••• |

Note: The number and the proportion of subjects for any protocol violation are reported

The denominator for calculating the proportions is the number of subjects in each analysis set

Source: Listing 16.2.2.1 - Protocol deviations

 $Program: Tables \backslash k345\text{-}dv\text{-}tbl.sas$ 



Table 14.2.1.1 - Total DF 2156Y concentrations (µg/mL) measured in plasma - PK Set 1

**Investigational Medicinal Product: Ladarixin fed (T)** 

| Statistics | Pre<br>dose | 0.25 h | 0.5 h | 1 h | 1.5 h | 2 h | 3 h | 4 h | 5 h | 6 h | 8 h | 10 h | 12 h | 18 h | 24 h | 30 h | 36 h | 48 h | 54 h | 60 h | 72 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| N | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| Geo.Mean | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | XXX.XX |
| Mean | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | XXX.XX |
| SD | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | XXX.XX |
| CV% | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | XXX.XX |
| Min | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | xxx.x | XXX.X | XXX.X | XXX.X | XXX.X | xxx.x | XXX.X | XXX.X | xxx.x | XXX.X | XXX.X |
| Median | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | XXX.XX |
| Max | XXX.X | XXX.X | xxx.x | xxx.x | XXX.X | xxx.x | XXX.X | xxx.x | xxx.x | XXX.X | xxx.x | xxx.x | xxx.x | xxx.x | XXX.X | XXX.X | xxx.x | xxx.x | XXX.X | xxx.x | XXX.X |

BLQL: Below Lower Quantification Limit (x.xx µg/mL)

Source: Listing 16.2.5.4 - Total DF 2156Y concentrations ( $\mu g/mL$ ) measured in plasma

 $Program: pk-analysis \verb|\k345-tlf.sas|$ 



Table 14.2.1.1 - Total DF 2156Y concentrations (µg/mL) measured in plasma - PK Set 1

**Investigational Medicinal Product: Ladarixin fasting (R)** 

| Statistics | Pre<br>dose | 0.25 h | 0.5 h | 1 h | 1.5 h | 2 h | 3 h | 4 h | 5 h | 6 h | 8 h | 10 h | 12 h | 18 h | 24 h | 30 h | 36 h | 48 h | 54 h | 60 h | 72 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| N | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| Geo.Mean | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | XXX.XX |
| Mean | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | XXX.XX |
| SD | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | XXX.XX |
| CV% | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | XXX.XX |
| Min | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | xxx.x | XXX.X | XXX.X | XXX.X | XXX.X | xxx.x | XXX.X | XXX.X | xxx.x | XXX.X | XXX.X |
| Median | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | XXX.XX |
| Max | XXX.X | XXX.X | xxx.x | xxx.x | XXX.X | xxx.x | XXX.X | xxx.x | xxx.x | XXX.X | xxx.x | xxx.x | xxx.x | xxx.x | XXX.X | XXX.X | xxx.x | xxx.x | XXX.X | xxx.x | XXX.X |

BLQL: Below Lower Quantification Limit (x.xx µg/mL)

Source: Listing 16.2.5.4 - Total DF 2156Y concentrations (µg/mL) measured in plasma

 $Program: pk-analysis \verb|\k345-tlf.sas|$ 



Table 14.2.1.2 - Unbound DF 2156Y concentrations (µg/mL) measured in plasma - PK Set 1

**Investigational Medicinal Product: Ladarixin fed (T)** 

| Statistics | 1 h | 3 h | 6 h | 12 h | 24 h |
|------------|--------|--------|--------|--------|--------|
| N | XX | XX | XX | XX | XX |
| Geo.Mean | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| Mean | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX |
| SD | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| CV% | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| Min | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |
| Median | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| Max | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |

BLQL: Below Lower Quantification Limit (x.xx µg/mL)

Source: Listing 16.2.5.5 - Unbound DF 2156Y concentrations (µg/mL) measured in plasma

Program: pk-analysis\k345-tlf.sas



Table 14.2.1.2 - Unbound DF 2156Y concentrations (µg/mL) measured in plasma - PK Set 1

**Investigational Medicinal Product: Ladarixin fasting (R)** 

| Statistics | 1 h | 3 h | 6 h | 12 h | 24 h |
|------------|--------|--------|--------|--------|--------|
| N | XX | XX | XX | XX | XX |
| Geo.Mean | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| Mean | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| SD | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| CV% | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| Min | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |
| Median | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| Max | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |

BLQL: Below Lower Quantification Limit (x.xx µg/mL)

Source: Listing 16.2.5.5 - Unbound DF 2156Y concentrations (µg/mL) measured in plasma

Program: pk-analysis\k345-tlf.sas



## Table 14.2.1.3 - DF 2108Y concentrations (µg/mL) measured in plasma - PK Set 2

**Investigational Medicinal Product: Ladarixin fed (T)** 

| Statistics | Pre<br>dose | 0.25 h | 0.5 h | 1 h | 1.5 h | 2 h | 3 h | 4 h | 5 h | 6 h | 8 h | 10 h | 12 h | 18 h | 24 h | 30 h | 36 h | 48 h | 54 h | 60 h | 72 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| N | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| Geo.Mean | XXX.XX | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | XXX.XX |
| Mean | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | XXX.XX |
| SD | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | XXX.XX |
| CV% | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | XXX.XX |
| Min | xxx.x | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | xxx.x | XXX.X | XXX.X | XXX.X | XXX.X |
| Median | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | XXX.XX |
| Max | XXX.X | XXX.X | XXX.X | XXX.X | xxx.x | xxx.x | xxx.x | XXX.X | XXX.X | XXX.X | XXX.X | xxx.x | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | xxx.x | XXX.X | XXX.X | XXX.X |

BLQL: Below Lower Quantification Limit (x.xx µg/mL)

Source: Listing 16.2.5.6 - DF 2108Y concentrations (μg/mL) measured in plasma

 $Program: pk-analysis \verb|\k345-tlf.sas|$ 



### Table 14.2.1.3 - DF 2108Y concentrations (µg/mL) measured in plasma - PK Set 2

**Investigational Medicinal Product: Ladarixin fasting (R)** 

| Statistics | | 0.25 h | 0.5 h | 1 h | 1.5 h | 2 h | 3 h | 4 h | 5 h | 6 h | 8 h | 10 h | 12 h | 18 h | 24 h | 30 h | 36 h | 48 h | 54 h | 60 h | 72 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | dose | | | | | | | | | | | | | | | | | | | | |
| N | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| Geo.Mean | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | XXX.XX |
| Mean | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | XXX.XX |
| SD | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | XXX.XX |
| CV% | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | XXX.XX |
| Min | XXX.X | XXX.X | xxx.x | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |
| Median | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | XXX.XX |
| Max | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |

BLQL: Below Lower Quantification Limit (x.xx µg/mL)

Source: Listing 16.2.5.6 - DF 2108Y concentrations (μg/mL) measured in plasma

 $Program: pk-analysis \verb|\k345-tlf.sas|$ 



# Table 14.2.1.4 - DF 2227Y concentrations (μg/mL) measured in plasma - PK Set 2

**Investigational Medicinal Product: Ladarixin fed (T)** 

| Statistics | Pre<br>dose | 0.25 h | 0.5 h | 1 h | 1.5 h | 2 h | 3 h | 4 h | 5 h | 6 h | 8 h | 10 h | 12 h | 18 h | 24 h | 30 h | 36 h | 48 h | 54 h | 60 h | 72 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| N | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| Geo.Mean | XXX.XX | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | XXX.XX |
| Mean | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | XXX.XX |
| SD | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | XXX.XX |
| CV% | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | XXX.XX |
| Min | xxx.x | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | xxx.x | XXX.X | XXX.X | XXX.X | XXX.X |
| Median | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | XXX.XX |
| Max | XXX.X | XXX.X | XXX.X | XXX.X | xxx.x | xxx.x | xxx.x | XXX.X | XXX.X | XXX.X | XXX.X | xxx.x | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | xxx.x | XXX.X | XXX.X | XXX.X |

BLQL: Below Lower Quantification Limit (x.xx µg/mL)

Source: Listing 16.2.5.7 - DF 2227Y concentrations (μg/mL) measured in plasma

 $Program: pk-analysis \verb|\k345-tlf.sas|$ 



## Table 14.2.1.4 - DF 2227Y concentrations (μg/mL) measured in plasma - PK Set 2

**Investigational Medicinal Product: Ladarixin fasting (R)** 

| Statistics | Pre<br>dose | 0.25 h | 0.5 h | 1 h | 1.5 h | 2 h | 3 h | 4 h | 5 h | 6 h | 8 h | 10 h | 12 h | 18 h | 24 h | 30 h | 36 h | 48 h | 54 h | 60 h | 72 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| N | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| Geo.Mean | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | XXX.XX |
| Mean | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | XXX.XX |
| SD | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | XXX.XX |
| CV% | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | XXX.XX |
| Min | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | xxx.x | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | xxx.x | XXX.X | XXX.X |
| Median | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | XXX.XX |
| Max | XXX.X | XXX.X | xxx.x | XXX.X | XXX.X | XXX.X | XXX.X | xxx.x | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |

BLQL: Below Lower Quantification Limit (x.xx µg/mL)

Source: Listing 16.2.5.7 - DF 2227Y concentrations (μg/mL) measured in plasma

 $Program: pk-analysis \verb|\k345-tlf.sas|$ 



Table 14.2.2.1 - Total DF 2156Y plasma PK parameters - PK Set 1

Investigational Medicinal Product: Ladarixin fed (T)

| Sex | Statistics | C <sub>max</sub><br>(μg/mL) | t <sub>max</sub><br>(h) | AUC <sub>0-t</sub><br>(h*µg/mL) | AUC <sub>0-inf</sub><br>(h*μg/mL) | t½<br>(h) | $\lambda_z$ (1/h) |
|---|---|---|---|---|---|---|---|
| Males | N | XX | XX | XX | XX | XX | XX |
| | Geo.Mean | XXX.XXX | XXX.XXX | XXX.XXX | XXX.XXX | XXX.XXX | XXX.XXX |
| | Mean | xxx.xxx | xxx.xxx | XXX.XXX | xxx.xxx | xxx.xxx | xxx.xxx |
| | SD | xxx.xxx | xxx.xxx | XXX.XXX | xxx.xxx | xxx.xxx | xxx.xxx |
| | CV% | xxx.xxx | xxx.xxx | XXX.XXX | XXX.XXX | xxx.xxx | xxx.xxx |
| | Min | xxx.xx | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX |
| | Median | xxx.xxx | xxx.xxx | XXX.XXX | XXX.XXX | xxx.xxx | XXX.XXX |
| | Max | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX |
| Females | N | XX | XX | XX | XX | XX | XX |
| | Geo.Mean | xxx.xxx | xxx.xxx | XXX.XXX | XXX.XXX | xxx.xxx | XXX.XXX |
| | Mean | xxx.xxx | xxx.xxx | XXX.XXX | xxx.xxx | xxx.xxx | xxx.xxx |
| | SD | xxx.xxx | xxx.xxx | XXX.XXX | XXX.XXX | xxx.xxx | XXX.XXX |
| | CV% | xxx.xxx | xxx.xxx | XXX.XXX | XXX.XXX | xxx.xxx | XXX.XXX |
| | Min | xxx.xx | xxx.xx | XXX.XX | xxx.xx | xxx.xx | xxx.xx |
| | Median | xxx.xxx | xxx.xxx | XXX.XXX | xxx.xxx | xxx.xxx | xxx.xxx |
| | Max | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |

Source: Listing 16.2.6.1 - Total DF 2156Y plasma PK parameters

Program: pk-analysis\k345-tlf.sas




Table 14.2.2.1 - Total DF 2156Y plasma PK parameters - PK Set 1

Investigational Medicinal Product: Ladarixin fed (T)

| Sex | Statistics | C <sub>max</sub><br>(μg/mL) | t <sub>max</sub><br>(h) | AUC <sub>0-t</sub><br>(h*μg/mL) | AUC <sub>0-inf</sub><br>(h*μg/mL) | t½<br>(h) | λ <sub>z</sub><br>(1/h) |
|---|---|---|---|---|---|---|---|
| Males and Females | N | XX | XX | XX | XX | XX | XX |
| | Geo.Mean | XXX.XXX | xxx.xxx | XXX.XXX | XXX.XXX | xxx.xxx | XXX.XXX |
| | Mean | XXX.XXX | xxx.xxx | XXX.XXX | XXX.XXX | xxx.xxx | XXX.XXX |
| | SD | XXX.XXX | xxx.xxx | XXX.XXX | XXX.XXX | XXX.XXX | XXX.XXX |
| | CV% | XXX.XXX | xxx.xxx | XXX.XXX | XXX.XXX | XXX.XXX | XXX.XXX |
| | Min | XXX.XX | xxx.xx | XXX.XX | XXX.XX | xxx.xx | XXX.XX |
| | Median | XXX.XXX | xxx.xxx | XXX.XXX | XXX.XXX | xxx.xxx | XXX.XXX |
| | Max | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |

Source: Listing 16.2.6.1 - Total DF 2156Y plasma PK parameters

Program: pk-analysis\k345-tlf.sas



Table 14.2.2.1 - Total DF 2156Y plasma PK parameters - PK Set 1

Investigational Medicinal Product: Ladarixin fasting (R)

| Sex | Statistics | C <sub>max</sub><br>(μg/mL) | t <sub>max</sub><br>(h) | AUC <sub>0-t</sub><br>(h*µg/mL) | AUC <sub>0-inf</sub><br>(h*μg/mL) | t½<br>(h) | $\lambda_z$ (1/h) |
|---|---|---|---|---|---|---|---|
| Males | N | XX | XX | XX | XX | XX | XX |
| | Geo.Mean | XXX.XXX | XXX.XXX | XXX.XXX | XXX.XXX | XXX.XXX | XXX.XXX |
| | Mean | xxx.xxx | xxx.xxx | XXX.XXX | xxx.xxx | xxx.xxx | xxx.xxx |
| | SD | xxx.xxx | xxx.xxx | XXX.XXX | xxx.xxx | xxx.xxx | xxx.xxx |
| | CV% | xxx.xxx | xxx.xxx | XXX.XXX | XXX.XXX | xxx.xxx | xxx.xxx |
| | Min | xxx.xx | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX |
| | Median | xxx.xxx | xxx.xxx | XXX.XXX | XXX.XXX | xxx.xxx | XXX.XXX |
| | Max | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX |
| Females | N | XX | XX | XX | XX | XX | XX |
| | Geo.Mean | xxx.xxx | xxx.xxx | XXX.XXX | XXX.XXX | xxx.xxx | XXX.XXX |
| | Mean | xxx.xxx | xxx.xxx | XXX.XXX | xxx.xxx | xxx.xxx | xxx.xxx |
| | SD | xxx.xxx | xxx.xxx | XXX.XXX | XXX.XXX | xxx.xxx | XXX.XXX |
| | CV% | xxx.xxx | xxx.xxx | XXX.XXX | XXX.XXX | xxx.xxx | XXX.XXX |
| | Min | xxx.xx | xxx.xx | XXX.XX | xxx.xx | xxx.xx | xxx.xx |
| | Median | xxx.xxx | xxx.xxx | XXX.XXX | xxx.xxx | xxx.xxx | xxx.xxx |
| | Max | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |

Source: Listing 16.2.6.1 - Total DF 2156Y plasma PK parameters

Program: pk-analysis\k345-tlf.sas



Table 14.2.2.1 - Total DF 2156Y plasma PK parameters - PK Set 1

Investigational Medicinal Product: Ladarixin fasting (R)

| Sex | Statistics | C <sub>max</sub><br>(μg/mL) | t <sub>max</sub><br>(h) | AUC <sub>0-t</sub><br>(h*μg/mL) | AUC <sub>0-inf</sub><br>(h*μg/mL) | t½<br>(h) | λ <sub>z</sub><br>(1/h) |
|---|---|---|---|---|---|---|---|
| Males and Females | N | XX | XX | XX | XX | XX | XX |
| | Geo.Mean | XXX.XXX | XXX.XXX | XXX.XXX | XXX.XXX | XXX.XXX | XXX.XXX |
| | Mean | xxx.xxx | xxx.xxx | XXX.XXX | xxx.xxx | xxx.xxx | xxx.xxx |
| | SD | xxx.xxx | xxx.xxx | XXX.XXX | xxx.xxx | xxx.xxx | xxx.xxx |
| | CV% | xxx.xxx | xxx.xxx | XXX.XXX | xxx.xxx | xxx.xxx | xxx.xxx |
| | Min | XXX.XX | xxx.xx | XXX.XX | XXX.XX | xxx.xx | XXX.XX |
| | Median | xxx.xxx | xxx.xxx | XXX.XXX | xxx.xxx | xxx.xxx | xxx.xxx |
| | Max | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |

Source: Listing 16.2.6.1 - Total DF 2156Y plasma PK parameters

Program: pk-analysis\k345-tlf.sas



Table 14.2.2.2 - DF 2108Y plasma PK parameters - PK Set 2

Investigational Medicinal Product: Ladarixin fed (T)

| Sex | Statistics | C <sub>max</sub><br>(μg/mL) | t <sub>max</sub><br>(h) | AUC <sub>0-t</sub><br>(h*μg/mL) | AUC <sub>0-inf</sub><br>(h*μg/mL) | t½<br>(h) | • <sub>z</sub> (1/h) |
|---|---|---|---|---|---|---|---|
| Males | N | XX | XX | XX | XX | XX | XX |
| | Geo.Mean | XXX.XXX | XXX.XXX | XXX.XXX | XXX.XXX | XXX.XXX | XXX.XXX |
| | Mean | XXX.XXX | XXX.XXX | XXX.XXX | XXX.XXX | XXX.XXX | XXX.XXX |
| | SD | xxx.xxx | xxx.xxx | XXX.XXX | XXX.XXX | xxx.xxx | XXX.XXX |
| | CV% | XXX.XXX | xxx.xxx | xxx.xxx | XXX.XXX | xxx.xxx | XXX.XXX |
| | Min | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| | Median | XXX.XXX | xxx.xxx | XXX.XXX | XXX.XXX | xxx.xxx | XXX.XXX |
| | Max | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | xxx.xx |
| Females | N | XX | xx | XX | XX | xx | XX |
| | Geo.Mean | XXX.XXX | xxx.xxx | xxx.xxx | XXX.XXX | xxx.xxx | xxx.xxx |
| | Mean | XXX.XXX | xxx.xxx | XXX.XXX | XXX.XXX | xxx.xxx | XXX.XXX |
| | SD | XXX.XXX | xxx.xxx | XXX.XXX | XXX.XXX | xxx.xxx | XXX.XXX |
| | CV% | XXX.XXX | xxx.xxx | XXX.XXX | XXX.XXX | xxx.xxx | xxx.xxx |
| | Min | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| | Median | XXX.XXX | xxx.xxx | XXX.XXX | XXX.XXX | xxx.xxx | xxx.xxx |
| | Max | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | xxx.xx |

Source: Listing 16.2.6.2 - DF 2108Y plasma PK parameters

Program: pk-analysis\k345-tlf.sas




# Table 14.2.2.2 - DF 2108Y plasma PK parameters - PK Set 2

Investigational Medicinal Product: Ladarixin fed (T)

| Sex | Statistics | C <sub>max</sub><br>(μg/mL) | t <sub>max</sub><br>(h) | AUC <sub>0-t</sub><br>(h*μg/mL) | AUC <sub>0-inf</sub><br>(h*μg/mL) | t½<br>(h) | • z<br>(1/h) |
|---|---|---|---|---|---|---|---|
| Males and Females | N | XX | XX | XX | XX | XX | XX |
| | Geo.Mean | XXX.XXX | xxx.xxx | XXX.XXX | XXX.XXX | XXX.XXX | XXX.XXX |
| | Mean | XXX.XXX | xxx.xxx | XXX.XXX | XXX.XXX | xxx.xxx | xxx.xxx |
| | SD | XXX.XXX | xxx.xxx | XXX.XXX | XXX.XXX | xxx.xxx | xxx.xxx |
| | CV% | XXX.XXX | xxx.xxx | XXX.XXX | XXX.XXX | xxx.xxx | XXX.XXX |
| | Min | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | xxx.xx |
| | Median | XXX.XXX | XXX.XXX | XXX.XXX | XXX.XXX | xxx.xxx | xxx.xxx |
| | Max | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |

Source: Listing 16.2.6.2 - DF 2108Y plasma PK parameters

Program: pk-analysis\k345-tlf.sas



Table 14.2.2.2 - DF 2108Y plasma PK parameters - PK Set 2

Investigational Medicinal Product: Ladarixin fasting (R)

| Sex | Statistics | C <sub>max</sub><br>(µg/mL) | t <sub>max</sub><br>(h) | AUC₀₁<br>(h*μg/mL) | AUC <sub>0-inf</sub><br>(h*µg/mL) | t½<br>(h) | • <sub>z</sub> (1/h) |
|---|---|---|---|---|---|---|---|
| Males | N | XX | XX | XX | XX | XX | XX |
| | Geo.Mean | XXX.XXX | XXX.XXX | XXX.XXX | XXX.XXX | XXX.XXX | XXX.XXX |
| | Mean | XXX.XXX | XXX.XXX | XXX.XXX | XXX.XXX | xxx.xxx | XXX.XXX |
| | SD | XXX.XXX | xxx.xxx | XXX.XXX | XXX.XXX | XXX.XXX | XXX.XXX |
| | CV% | xxx.xxx | xxx.xxx | XXX.XXX | XXX.XXX | XXX.XXX | XXX.XXX |
| | Min | XXX.XX | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx |
| | Median | XXX.XXX | xxx.xxx | XXX.XXX | XXX.XXX | xxx.xxx | xxx.xxx |
| | Max | XXX.XX | xxx.xx | XXX.XX | XXX.XX | xxx.xx | XXX.XX |
| Females | N | XX | XX | XX | XX | XX | XX |
| | Geo.Mean | xxx.xxx | xxx.xxx | XXX.XXX | XXX.XXX | xxx.xxx | XXX.XXX |
| | Mean | xxx.xxx | xxx.xxx | XXX.XXX | XXX.XXX | XXX.XXX | XXX.XXX |
| | SD | xxx.xxx | xxx.xxx | XXX.XXX | XXX.XXX | XXX.XXX | XXX.XXX |
| | CV% | xxx.xxx | xxx.xxx | XXX.XXX | XXX.XXX | XXX.XXX | XXX.XXX |
| | Min | XXX.XX | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX |
| | Median | XXX.XXX | xxx.xxx | xxx.xxx | xxx.xxx | xxx.xxx | xxx.xxx |
| | Max | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |

Source: Listing 16.2.6.2 - DF 2108Y plasma PK parameters

Program: pk-analysis\k345-tlf.sas



Table 14.2.2.2 - DF 2108Y plasma PK parameters - PK Set 2

Investigational Medicinal Product: Ladarixin fasting (R)

| Sex | Statistics | C <sub>max</sub><br>(μg/mL) | t <sub>max</sub><br>(h) | AUC <sub>0-t</sub><br>(h*μg/mL) | AUC <sub>0-inf</sub><br>(h*μg/mL) | t½<br>(h) | • z<br>(1/h) |
|---|---|---|---|---|---|---|---|
| Males and Females | N | XX | XX | XX | XX | XX | XX |
| | Geo.Mean | XXX.XXX | xxx.xxx | XXX.XXX | XXX.XXX | XXX.XXX | XXX.XXX |
| | Mean | XXX.XXX | xxx.xxx | XXX.XXX | XXX.XXX | xxx.xxx | xxx.xxx |
| | SD | XXX.XXX | xxx.xxx | XXX.XXX | XXX.XXX | xxx.xxx | xxx.xxx |
| | CV% | XXX.XXX | xxx.xxx | XXX.XXX | XXX.XXX | xxx.xxx | XXX.XXX |
| | Min | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | xxx.xx |
| | Median | XXX.XXX | XXX.XXX | XXX.XXX | XXX.XXX | xxx.xxx | xxx.xxx |
| | Max | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |

Source: Listing 16.2.6.2 - DF 2108Y plasma PK parameters

Program: pk-analysis\k345-tlf.sas



Table 14.2.2.3 - DF 2227Y plasma PK parameters - PK Set 2

Investigational Medicinal Product: Ladarixin fed (T)

| Sex | Statistics | C <sub>max</sub><br>(μg/mL) | t <sub>max</sub><br>(h) | AUC <sub>0-t</sub><br>(h*μg/mL) | AUC <sub>0-inf</sub><br>(h*μg/mL) | t½<br>(h) | • <sub>z</sub> (1/h) |
|---|---|---|---|---|---|---|---|
| Males | N | XX | XX | XX | XX | XX | XX |
| | Geo.Mean | XXX.XXX | XXX.XXX | XXX.XXX | XXX.XXX | XXX.XXX | XXX.XXX |
| | Mean | XXX.XXX | xxx.xxx | XXX.XXX | XXX.XXX | xxx.xxx | XXX.XXX |
| | SD | XXX.XXX | xxx.xxx | xxx.xxx | xxx.xxx | xxx.xxx | XXX.XXX |
| | CV% | XXX.XXX | xxx.xxx | xxx.xxx | xxx.xxx | xxx.xxx | XXX.XXX |
| | Min | xxx.xx | xxx.xx | XXX.XX | XXX.XX | xxx.xx | XXX.XX |
| | Median | XXX.XXX | xxx.xxx | XXX.XXX | XXX.XXX | xxx.xxx | XXX.XXX |
| | Max | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | xxx.xx |
| Females | N | XX | XX | XX | XX | XX | XX |
| | Geo.Mean | XXX.XXX | xxx.xxx | xxx.xxx | xxx.xxx | xxx.xxx | xxx.xxx |
| | Mean | XXX.XXX | xxx.xxx | xxx.xxx | xxx.xxx | xxx.xxx | XXX.XXX |
| | SD | XXX.XXX | xxx.xxx | XXX.XXX | XXX.XXX | xxx.xxx | XXX.XXX |
| | CV% | XXX.XXX | xxx.xxx | XXX.XXX | XXX.XXX | xxx.xxx | xxx.xxx |
| | Min | XXX.XX | xxx.xx | XXX.XX | XXX.XX | xxx.xx | XXX.XX |
| | Median | XXX.XXX | xxx.xxx | XXX.XXX | XXX.XXX | xxx.xxx | xxx.xxx |
| | Max | XXX.XX | xxx.xx | XXX.XX | XXX.XX | xxx.xx | XXX.XX |

Source: Listing 16.2.6.3 - DF 2227Y plasma PK parameters

Program: pk-analysis\k345-tlf.sas




Table 14.2.2.3 - DF 2227Y plasma PK parameters - PK Set 2

Investigational Medicinal Product: Ladarixin fed (T)

| Sex | Statistics | C <sub>max</sub><br>(μg/mL) | t <sub>max</sub><br>(h) | AUC <sub>0-t</sub><br>(h*μg/mL) | AUC <sub>0-inf</sub><br>(h*μg/mL) | t½<br>(h) | • z<br>(1/h) |
|---|---|---|---|---|---|---|---|
| Males and Females | N | XX | XX | XX | XX | XX | XX |
| | Geo.Mean | XXX.XXX | xxx.xxx | XXX.XXX | XXX.XXX | XXX.XXX | XXX.XXX |
| | Mean | XXX.XXX | xxx.xxx | XXX.XXX | XXX.XXX | xxx.xxx | xxx.xxx |
| | SD | XXX.XXX | xxx.xxx | XXX.XXX | XXX.XXX | xxx.xxx | xxx.xxx |
| | CV% | XXX.XXX | xxx.xxx | XXX.XXX | XXX.XXX | xxx.xxx | xxx.xxx |
| | Min | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | xxx.xx |
| | Median | XXX.XXX | XXX.XXX | XXX.XXX | XXX.XXX | xxx.xxx | xxx.xxx |
| | Max | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |

Source: Listing 16.2.6.3 - DF 2227Y plasma PK parameters

Program: pk-analysis\k345-tlf.sas



Table 14.2.2.3 - DF 2227Y plasma PK parameters - PK Set 2

Investigational Medicinal Product: Ladarixin fasting (R)

| Sex | Statistics | C <sub>max</sub><br>(μg/mL) | t <sub>max</sub><br>(h) | AUC₀₁<br>(h*μg/mL) | AUC <sub>0-inf</sub><br>(h*µg/mL) | t½<br>(h) | • <sub>z</sub> (1/h) |
|---|---|---|---|---|---|---|---|
| | | | | | | | _ |
| Males | N | XX | XX | XX | XX | XX | XX |
| | Geo.Mean | XXX.XXX | XXX.XXX | XXX.XXX | XXX.XXX | XXX.XXX | XXX.XXX |
| | Mean | xxx.xxx | xxx.xxx | XXX.XXX | xxx.xxx | xxx.xxx | xxx.xxx |
| | SD | xxx.xxx | xxx.xxx | XXX.XXX | XXX.XXX | xxx.xxx | xxx.xxx |
| | CV% | xxx.xxx | xxx.xxx | XXX.XXX | XXX.XXX | xxx.xxx | xxx.xxx |
| | Min | xxx.xx | XXX.XX | XXX.XX | XXX.XX | xxx.xx | xxx.xx |
| | Median | xxx.xxx | xxx.xxx | XXX.XXX | XXX.XXX | xxx.xxx | xxx.xxx |
| | Max | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | xxx.xx |
| Females | N | XX | XX | XX | XX | XX | XX |
| | Geo.Mean | xxx.xxx | xxx.xxx | XXX.XXX | XXX.XXX | xxx.xxx | xxx.xxx |
| | Mean | xxx.xxx | xxx.xxx | XXX.XXX | XXX.XXX | xxx.xxx | xxx.xxx |
| | SD | xxx.xxx | xxx.xxx | XXX.XXX | XXX.XXX | XXX.XXX | xxx.xxx |
| | CV% | XXX.XXX | xxx.xxx | XXX.XXX | XXX.XXX | XXX.XXX | XXX.XXX |
| | Min | xxx.xx | xxx.xx | XXX.XX | xxx.xx | XXX.XX | xxx.xx |
| | Median | xxx.xxx | xxx.xxx | XXX.XXX | XXX.XXX | xxx.xxx | xxx.xxx |
| | Max | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |

Source: Listing 16.2.6.3 - DF 2227Y plasma PK parameters

Program: pk-analysis\k345-tlf.sas



Table 14.2.2.3 - DF 2227Y plasma PK parameters - PK Set 2

Investigational Medicinal Product: Ladarixin fasting (R)

| Sex | Statistics | C <sub>max</sub><br>(μg/mL) | t <sub>max</sub><br>(h) | AUC <sub>0-t</sub><br>(h*µg/mL) | AUC <sub>0-inf</sub><br>(h*μg/mL) | t½<br>(h) | • z<br>(1/h) |
|---|---|---|---|---|---|---|---|
| Males and Females | N | XX | XX | XX | XX | XX | XX |
| | Geo.Mean | XXX.XXX | XXX.XXX | XXX.XXX | XXX.XXX | XXX.XXX | XXX.XXX |
| | Mean | XXX.XXX | XXX.XXX | XXX.XXX | XXX.XXX | XXX.XXX | XXX.XXX |
| | SD | XXX.XXX | xxx.xxx | XXX.XXX | XXX.XXX | xxx.xxx | xxx.xxx |
| | CV% | XXX.XXX | XXX.XXX | XXX.XXX | XXX.XXX | XXX.XXX | XXX.XXX |
| | Min | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| | Median | XXX.XXX | XXX.XXX | XXX.XXX | XXX.XXX | XXX.XXX | XXX.XXX |
| | Max | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |

Source: Listing 16.2.6.3 - DF 2227Y plasma PK parameters

Program: pk-analysis\k345-tlf.sas



Table 14.2.2.4 - Total DF 2156Y, DF 2108Y and DF 2227Y relative bioavailability in plasma calculated as AUC<sub>0-t</sub> T/R ratio - PK Sets 1 and 2

| Sex | Statistics | DF 2156Y Frel <sup>1</sup> (%) | DF 2108Y Frel <sup>2</sup> (%) | DF 2227Y Fret <sup>2</sup> (%) |
|---|---|---|---|---|
| Males | N | XX | XX | XX |
| | Geo.Mean | XXX.XXX | XXX.XXX | XXX.XXX |
| | Mean | XXX.XXX | xxx.xxx | xxx.xxx |
| | SD | XXX.XXX | xxx.xxx | xxx.xxx |
| | CV% | XXX.XXX | xxx.xxx | xxx.xxx |
| | Min | xxx.xx | xxx.xx | xxx.xx |
| | Median | XXX.XXX | xxx.xxx | xxx.xxx |
| | Max | XXX.XX | XXX.XX | XXX.XX |
| Females | N | XX | XX | xx |
| | Geo.Mean | xxx.xxx | xxx.xxx | xxx.xxx |
| | Mean | xxx.xxx | xxx.xxx | xxx.xxx |
| | SD | xxx.xxx | xxx.xxx | xxx.xxx |
| | CV% | xxx.xxx | xxx.xxx | xxx.xxx |
| | Min | xxx.xx | xxx.xx | xxx.xx |
| | Median | xxx.xxx | XXX.XXX | XXX.XXX |
| | Max | xxx.xx | XXX.XX | XXX.XX |

T: Ladarixin fed (T)

R: Ladarixin fasting (R)

Note 1: PK set 1 Note 2: PK set 2

Source: Listing 16.2.6.4 - Total DF 2156Y, DF 2108Y and DF 2227Y relative bioavailability in plasma calculated as AUC<sub>0-t</sub> T/R ratio

Program: pk-analysis\k345-tlf.sas



Table 14.2.2.4 - Total DF 2156Y, DF 2108Y and DF 2227Y relative bioavailability in plasma calculated as AUC<sub>0-t</sub> T/R ratio - PK Sets 1 and 2

| Sex | Statistics | DF 2156Y Frel <sup>1</sup> (%) | DF 2108Y Fret <sup>2</sup> (%) | DF 2227Y Frel <sup>2</sup> (%) |
|---|---|---|---|---|
| Males and Females | N | XX | xx | xx |
| | Geo.Mean | xxx.xxx | xxx.xxx | xxx.xxx |
| | Mean | xxx.xxx | xxx.xxx | xxx.xxx |
| | SD | xxx.xxx | xxx.xxx | xxx.xxx |
| | CV% | xxx.xxx | xxx.xxx | xxx.xxx |
| | Min | xxx.xx | xxx.xx | xxx.xx |
| | Median | XXX.XXX | XXX.XXX | XXX.XXX |
| | Max | XXX.XX | XXX.XX | XXX.XX |

T: Ladarixin fed (T)
R: Ladarixin fasting (R)

Note 1: PK set 1 Note 2: PK set 2

Source: Listing 16.2.6.4 - Total DF 2156Y, DF 2108Y and DF 2227Y relative bioavailability in plasma calculated as AUC<sub>0-t</sub> T/R ratio

Program: pk-analysis\k345-tlf.sas



Table 14.2.3.1 - Statistical analysis on total DF 2156Y plasma PK parameters - PK set 1

| Analysis | Dependent Variable | Comparison | Point Estimate | 90% Confidence Interval<br>Lower Limit | 90% Confidence Interval<br>Upper Limit | Effect | p Value |
|---|---|---|---|---|---|---|---|
| ANOVA | $Ln(AUC_{0-inf})$ | T vs R | XXX.XX | XXX.XX | XXX.XX | | |
| | ( 0-mi) | | | | | Sequence | X.XXXX |
| | | | | | | Treatment | x.xxxx |
| | | | | | | Period | x.xxxx |
| ANOVA | $Ln(AUC_{0-1})$ | T vs R | XXX.XX | XXX.XX | XXX.XX | | |
| | | | | | | Sequence | XXXXX |
| | | | | | | Treatment | X.XXXX |
| | | | | | | Period | X.XXXX |
| ANOVA | $Ln(C_{max})$ | T vs R | XXX.XX | XXX.XX | XXX.XX | | |
| | | | | | | Sequence | X.XXXX |
| | | | | | | Treatment | X.XXXX |
| | | | | | | Period | x.xxxx |

T: Ladarixin fed (T)

R: Ladarixin fasting (R)

Program: pk-analysis\k345-tlf.sas



Table 14.2.3.2 - Statistical analysis of gender effect on total DF 2156Y plasma PK parameters - PK set 1

| Analysis | Treatment | Dependent Variable | Comparison | p Value |
|---|---|---|---|---|
| Wilcoxon | Ladarixin fed (T) | $\mathrm{AUC}_{0	ext{-}\mathrm{inf}}$ | Males vs Females | x.xxxx |
| WILCOXOII | Laudiixiii icu (1) | $\mathrm{AUC}_{0	ext{-inf}}$ | Males vs Females | X.XXXX |
| | | $C_{max}$ | Males vs Females | X.XXXX |
| Wilcoxon | Ladarixin fasting (R) | $\mathrm{AUC}_{0	ext{-inf}}$ | Males vs Females | X.XXXX |
| | | $\mathrm{AUC}_{0	ext{-t}}$ | Males vs Females | X.XXXX |
| | | $C_{max}$ | Males vs Females | X.XXXX |

Program: pk-analysis\k345-tlf.sas



Table 14.2.3.3 - Statistical analysis of gender effect on DF 2108Y plasma PK parameters - PK set 2

| Analysis | Treatment | Dependent Variable | Comparison | p Value |
|---|---|---|---|---|
| Wilcoxon | Ladarixin fed (T) | $\mathrm{AUC}_{0	ext{-inf}}$ | Males vs Females | V VVVV |
| WIICOXOII | Ladarixiii led (1) | $\mathrm{AUC}_{0	ext{-inf}}$ | Males vs Females | X,XXXX<br>X,XXXX |
| | | $C_{\max}$ | Males vs Females | X.XXXX |
| Wilcoxon | Ladarixin fasting (R) | $\mathrm{AUC}_{0	ext{-inf}}$ | Males vs Females | X.XXXX |
| | | $\mathrm{AUC}_{0	ext{-t}}$ | Males vs Females | X.XXXX |
| | | $C_{max}$ | Males vs Females | X.XXXX |

Program: pk-analysis\k345-tlf.sas



Table 14.2.3.4 - Statistical analysis of gender effect on DF 2227Y plasma PK parameters - PK set 2

| Analysis | Treatment | Dependent Variable | Comparison | p Value |
|---|---|---|---|---|
| Wilcoxon | Ladarixin fed (T) | $\begin{array}{c} AUC_{0\text{-}\mathrm{inf}} \\ AUC_{0\text{-}\mathrm{t}} \\ C_{max} \end{array}$ | Males vs Females<br>Males vs Females<br>Males vs Females | X.XXXX<br>X.XXXX<br>X.XXXX |
| Wilcoxon | Ladarixin fasting (R) | $egin{array}{l} { m AUC_{0-inf}} \ { m AUC_{0-t}} \ { m C_{max}} \end{array}$ | Males vs Females<br>Males vs Females<br>Males vs Females | X.XXXX<br>X.XXXX<br>X.XXXX |

Program: pk-analysis\k345-tlf.sas



Table 14.3.1.1 - Global incidence of subjects with treatment-emergent adverse events - Safety set

| | Ladarixin<br>fed (T)<br>N=XX<br>n (%) [n AE] | Safety Set Ladarixin fasting (R) N=XX n (%) [n AE] | Overall<br>N=XX<br>n (%) [n AE] |
|---|---|---|---|
| Treatment-emergent Adverse Events | nn (xx.x) [kk] | nn(xx.x)[kk] | nn(xx.x)[kk] |
| Relationship | nn (xx.x) [kk] | nn (xx.x) [kk] | nn (xx.x) [kk] |
| Related | nn(xx.x)[kk] | nn(xx.x)[kk] | nn(xx.x)[kk] |
| Not related | $\operatorname{nn}(xx.x)[kk]$ | nn(xx.x)[kk] | nn(xx.x)[kk] |
| Intensity | nn (xx.x) [kk] | nn (xx.x) [kk] | nn (xx.x) [kk] |
| Mild | nn(xx.x)[kk] | nn(xx.x)[kk] | nn(xx.x)[kk] |
| Moderate | nn(xx.x)[kk] | nn(xx.x)[kk] | nn(xx.x)[kk] |
| Severe | nn (xx.x) [kk] | nn(xx.x)[kk] | nn(xx.x)[kk] |
| Leading to discontinuation | nn(xx.x)[kk] | nn(xx.x)[kk] | nn(xx.x)[kk] |

Note: Subjects are summarised according to the product they actually received

Subjects are summarised according to the each level of relationship and intensity reported in each treatment group and overall

The number and the proportion of subjects with any adverse event and the number of adverse events for each classification level are reported

The denominator for calculating the proportions is the number of subjects in the safety set of each treatment group and overall

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

 $Program: Tables \verb|\k345-ae-01-tbl.sas|$ 



Table 14.3.1.1 - Global incidence of subjects with treatment-emergent adverse events - Safety set

| | Ladarixin<br>fed (T)<br>N=XX<br>n (%) [n AE] | Safety Set Ladarixin fasting (R) N=XX n (%) [n AE] | Overall<br>N=XX<br>n (%) [n AE] |
|---|---|---|---|
| Serious Treatment-emergent Adverse Events | nn(xx.x)[kk] | nn(xx.x)[kk] | nn(xx.x)[kk] |
| Relationship | nn(xx.x)[kk] | nn (xx.x) [kk] | nn(xx.x)[kk] |
| Related | nn(xx.x)[kk] | nn(xx.x)[kk] | nn(xx.x)[kk] |
| Not related | $\operatorname{nn}(xx.x)[kk]$ | nn(xx.x)[kk] | nn(xx.x)[kk] |
| Intensity | nn (xx.x) [kk] | nn (xx.x) [kk] | nn (xx.x) [kk] |
| Mild | nn(xx.x)[kk] | nn(xx.x)[kk] | nn(xx.x)[kk] |
| Moderate | nn(xx.x)[kk] | nn(xx.x)[kk] | nn(xx.x)[kk] |
| Severe | nn(xx.x)[kk] | nn(xx.x)[kk] | nn(xx.x)[kk] |
| Leading to discontinuation | nn(xx.x)[kk] | nn(xx.x)[kk] | nn(xx.x)[kk] |

Note: Subjects are summarised according to the product they actually received

Subjects are summarised according to the each level of relationship and intensity reported in each treatment group and overall

The number and the proportion of subjects with any adverse event and the number of adverse events for each classification level are reported

The denominator for calculating the proportions is the number of subjects in the safety set of each treatment group and overall

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k345-ae-01-tbl.sas



Table 14.3.1.2 - Subjects with treatment-emergent adverse events by system organ class and preferred term - Safety set

| | Safety Set | | |
|---|---|---|---|
| System Organ Class <sup>1</sup> Preferred Term <sup>1</sup> | Ladarixin<br>fed (T)<br>N=XX<br>n (%) [n AE] | Ladarixin<br>fasting (R)<br>N=XX<br>n (%) [n AE] | Overall<br>N=XX<br>n (%) [n AE] |
| Treatment-emergent Adverse Events | nn(xx.x)[kk] | nn (xx.x) [kk] | nn (xx.x) [kk] |
| Nervous system disorders | nn(xx.x)[kk] | nn (xx.x) [kk] | nn(xx.x)[kk] |
| Headache | nn (xx.x) [kk] | nn (xx.x) [kk] | nn (xx.x) [kk] |
| Gastrointestinal disorders | nn(xx.x)[kk] | nn (xx.x) [kk] | nn(xx.x)[kk] |
| Abdominal pain upper<br>Diarrhoea | nn(xx.x)[kk] $nn(xx.x)[kk]$ | nn (xx.x) [kk]<br>nn (xx.x) [kk] | nn (xx.x) [kk]<br>nn (xx.x) [kk] |

Note: Subjects are summarised according to the product they actually received

The number and the proportion of subjects with any adverse event and the number of adverse events for each classification level are reported

The denominator for calculating the proportions is the number of subjects in the safety set of each treatment group and overall

Note 1: MedDRA version 23.1

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k345-ae-02-tbl.sas


Table 14.3.1.3 - Subjects with treatment-emergent adverse events by intensity, system organ class and preferred term - Safety set

| | Safety Set Ladarixin fed (T) N=XX Ladarixin fasting (R) N=XX | | | | | Overall<br>N=XX | | | |
|---|---|---|---|---|---|---|---|---|---|
| System Organ Class <sup>1</sup><br>Preferred Term <sup>1</sup> | Mild<br>n (%) [n AE] | Moderate<br>n (%) [n AE] | Severe<br>n (%) [n AE] | Mild<br>n (%) [n AE] | Moderate<br>n (%) [n AE] | Severe<br>n (%) [n AE] | Mild<br>n (%) [n AE] | Moderate<br>n (%) [n AE] | Severe<br>n (%) [n AE] |
| Treatment-emergent Adverse Events | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] |
| Nervous system disorders | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] |
| Headache | nn(x.x)[kk] $nn(x.x)[kk]$ | nn (x.x) [kk]<br>nn (x.x) [kk] | nn (x.x) [kk]<br>nn (x.x) [kk] | nn (x.x) [kk]<br>nn (x.x) [kk] | nn (x.x) [kk]<br>nn (x.x) [kk] | nn (x.x) [kk]<br>nn (x.x) [kk] | nn (x.x) [kk]<br>nn (x.x) [kk] | nn (x.x) [kk]<br>nn (x.x) [kk] | nn (x.x) [kk]<br>nn (x.x) [kk] |
| Gastrointestinal disorders | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] |
| Abdominal pain upper<br>Diarrhoea | nn (x.x) [kk]<br>nn (x.x) [kk]<br>nn (x.x) [kk] | nn (x.x) [kk]<br>nn (x.x) [kk]<br>nn (x.x) [kk] | nn (x.x) [kk]<br>nn (x.x) [kk]<br>nn (x.x) [kk] | nn (x.x) [kk]<br>nn (x.x) [kk]<br>nn (x.x) [kk] | nn (x.x) [kk]<br>nn (x.x) [kk]<br>nn (x.x) [kk] | nn (x.x) [kk]<br>nn (x.x) [kk]<br>nn (x.x) [kk] | nn (x.x) [kk]<br>nn (x.x) [kk]<br>nn (x.x) [kk] | nn (x.x) [kk]<br>nn (x.x) [kk]<br>nn (x.x) [kk] | nn (x.x) [kk]<br>nn (x.x) [kk]<br>nn (x.x) [kk] |

Note: Subjects are summarised according to the treatment they actually received

The number and the proportion of subjects with any adverse event and the number of adverse events for each classification level are reported

The denominator for calculating the proportions is the number of subjects in the safety set of each treatment group and overall

Note 1: MedDRA version 23.1

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k345-ae-02-tbl.sas




Table 14.3.1.4 - Subjects with treatment-emergent adverse events related to the IMP by system organ class and preferred term - Safety set

| | Safety Set | | |
|---|---|---|---|
| System Organ Class <sup>1</sup> Preferred Term <sup>1</sup> | Ladarixin<br>fed (T)<br>N=XX<br>n (%) [n AE] | Ladarixin<br>fasting (R)<br>N=XX<br>n (%) [n AE] | Overall<br>N=XX<br>n (%) [n AE] |
| Treatment-emergent Adverse Events related to the IMP | nn(xx.x)[kk] | nn (xx.x) [kk] | nn (xx.x) [kk] |
| Nervous system disorders | nn(xx.x)[kk] | nn (xx.x) [kk] | nn (xx.x) [kk] |
| Headache | nn(xx.x)[kk] | nn(xx.x)[kk] | nn(xx.x)[kk] |
| <del></del> | <del></del> | | |
| Gastrointestinal disorders | nn(xx.x)[kk] | nn(xx.x)[kk] | nn(xx.x)[kk] |
| Abdominal pain upper | nn(xx.x)[kk] | nn (xx.x) [kk] | nn (xx.x) [kk] |
| Diarrhoea | nn(xx.x)[kk] | nn(xx.x)[kk] | nn(xx.x)[kk] |
| <u></u> | | | |

Note: Subjects are summarised according to the product they actually received

The number and the proportion of subjects with any related adverse event and the number of related adverse events for each classification level are reported

The denominator for calculating the proportions is the number of subjects in the safety set of each treatment group and overall

Note 1: MedDRA version 23.1

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k345-ae-02-tbl.sas




Table 14.3.1.5 - Subjects with serious treatment-emergent adverse events by system organ class and preferred term - Safety set

| | Safety Set | | |
|---|---|---|---|
| System Organ Class <sup>1</sup> Preferred Term <sup>1</sup> | Ladarixin<br>fed (T)<br>N=XX<br>n (%) [n AE] | Ladarixin<br>fasting (R)<br>N=XX<br>n (%) [n AE] | Overall<br>N=XX<br>n (%) [n AE] |
| Serious Treatment-emergent Adverse Events | nn(xx.x)[kk] | nn (xx.x) [kk] | nn (xx.x) [kk] |
| Nervous system disorders | nn(xx.x)[kk] | nn (xx.x) [kk] | nn(xx.x)[kk] |
| Headache | nn (xx.x) [kk] | nn (xx.x) [kk]<br> | nn (xx.x) [kk] |
| Gastrointestinal disorders | nn (xx.x) [kk] | nn(xx.x)[kk] | nn (xx.x) [kk] |
| Abdominal pain upper<br>Diarrhoea | nn (xx.x) [kk]<br>nn (xx.x) [kk] | nn (xx.x) [kk]<br>nn (xx.x) [kk] | nn (xx.x) [kk]<br>nn (xx.x) [kk] |
| | ··· | ••• | ••• |

Note: Subjects are summarised according to the product they actually received

The number and the proportion of subjects with any serious adverse event and the number of serious adverse events for each classification level are reported

The denominator for calculating the proportions is the number of subjects in the safety set of each treatment group and overall

Note 1: MedDRA version 23.1

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k345-ae-02-tbl.sas



Table 14.3.1.6 - Subjects with serious treatment-emergent adverse events related to the IMP by system organ class and preferred term - Safety set

| | Safety Set | | |
|---|---|---|---|
| System Organ Class <sup>1</sup> Preferred Term <sup>1</sup> | Ladarixin<br>fed (T)<br>N=XX<br>n (%) [n AE] | Ladarixin<br>fasting (R)<br>N=XX<br>n (%) [n AE] | Overall<br>N=XX<br>n (%) [n AE] |
| Serious Treatment-emergent Adverse Events related to the IMP | nn (xx.x) [kk] | nn(xx.x)[kk] | nn (xx.x) [kk] |
| Nervous system disorders | nn(xx.x)[kk] | nn(xx.x)[kk] | nn(xx.x)[kk] |
| Headache | nn (xx.x) [kk] | nn (xx.x) [kk] | nn (xx.x) [kk] |
| Gastrointestinal disorders | nn (xx.x) [kk] | nn (xx.x) [kk] | nn (xx.x) [kk] |
| Abdominal pain upper<br>Diarrhoea | nn (xx.x) [kk]<br>nn (xx.x) [kk] | nn (xx.x) [kk]<br>nn (xx.x) [kk] | nn(xx.x)[kk] $nn(xx.x)[kk]$ |
| <br> | | ••• | |

Note: Subjects are summarised according to the product they actually received

The number and the proportion of subjects with any serious related adverse event and the number of serious related adverse events for each classification level are reported. The denominator for calculating the proportions is the number of subjects in the safety set of each treatment group and overall

Note 1: MedDRA version 23.1

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k345-ae-02-tbl.sas



Table 14.3.2.1 - Treatment emergent adverse events leading to death, serious adverse events or treatment emergent adverse events leading to discontinuation - Safety set

#### **Investigational Medicinal Product: Ladarixin fed (T)**

| Subject<br>ID | Adverse<br>Event<br>ID | Follow<br>Up<br>ID | | |
|---|---|---|---|---|
| S001/001 | 1 | | Description: | Headache |
| | | | Preferred Term <sup>1</sup> : | Headache |
| | | | System Organ Class <sup>1</sup> : | Nervous system disorders |
| | | | Start Date/Time - End Date/Time (Day): | ddMMMyyyy hh:mm (k) - ddMMMyyyy hh:mm (j) |
| | | | IMP last administration before AE onset Date and Time: | ddMMMyyyy hh:mm |
| | | | Time Elapsed form Last Study Drug intake before AE | hh:mm |
| | | | Relationship to Study Drug Treatment (IMP): | N |
| | | | Severity | Mild |
| | | | AE frequency | Intermittent |
| | | | Serious Adverse Event? | N |
| | | | Seriousness criteria: | |
| | | | Action Taken with Study Drug Treatment (IMP): | Dose not changed |
| | | | Any Concomitant Medication?: | Y |
| | | | Caused study discontinuation | Y |
| | | | Other Action Taken: | |
| | | | Outcome: | Recovered/Resolved |
| | | | Comments: | |

Note: Subjects are listed according to the product they actually received

Note 1: MedDRA version 23.1.

Sources: Listing 16.2.7.1 - Treatment-emergent adverse events, Listing 16.2.7.2 - Pre-treatment adverse events (for serious adverse events only)

Program: Tables\k345-ae-03-tbl.sas



Table 14.3.2.1 - Treatment emergent adverse events leading to death, serious adverse events or treatment emergent adverse events leading to discontinuation - Safety set

**Investigational Medicinal Product: Ladarixin fasting (R)** 

| Subject<br>ID | Adverse<br>Event<br>ID | Follow<br>Up<br>ID | | |
|---|---|---|---|---|
| S001/001 | 2 | | Description: | Headache |
| | | | Preferred Term <sup>1</sup> : | Headache |
| | | | System Organ Class <sup>1</sup> : | Nervous system disorders |
| | | | Start Date/Time - End Date/Time (Day): | ddMMMyyyy hh:mm (k) - ddMMMyyyy hh:mm (j) |
| | | | IMP last administration before AE onset Date and Time: | ddMMMyyyy hh:mm |
| | | | Time Elapsed form Last Study Drug intake before AE | hh:mm |
| | | | Relationship to Study Drug Treatment (IMP): | N |
| | | | Severity | Mild |
| | | | AE frequency | Intermittent |
| | | | Serious Adverse Event? | N |
| | | | Seriousness criteria: | |
| | | | Action Taken with Study Drug Treatment (IMP): | Dose not changed |
| | | | Any Concomitant Medication?: | Y |
| | | | Caused study discontinuation | Y |
| | | | Other Action Taken: | |
| | | | Outcome: | Recovered/Resolved |
| | | | Comments: | |
| ••• | ••• | | | |

Note: Subjects are listed according to the product they actually received

Note 1: MedDRA version 23.1.

Sources: Listing 16.2.7.1 - Treatment-emergent adverse events, Listing 16.2.7.2 - Pre-treatment adverse events (for serious adverse events only)

Program: Tables\k345-ae-03-tbl.sas



# Table 14.3.4.1 - Abnormal laboratory values - Safety set

**Category of Laboratory Parameters: BLOOD CHEMISTRY** 

| Subject | Time | Collection | Parameter | Value and | Normal Range or | Clinically |
|---|---|---|---|---|---|---|
| ID | Point | Date/time | | Abnormality <sup>1</sup> | Reference Value | Significant? |
| S001/001 | Screening | ddMMMyyyy hh:mm | Phosphate [mmol/L] | 0.84 [L] | 0.87 - 1.45 | N |
| S001/001 | | | | | | |
| | End of Study | ddMMMyyyy hh:mm | Phosphate [mmol/L] | 0.84 [L] | 0.87 - 1.45 | N |
| ••• | ••• | ••• | <del></del> | ••• | ••• | ••• |

Note 1: H=Higher than upper normal limit, L=Lower than lower normal limit

Source: Listing 16.2.8.1 - Individual laboratory measurements

Program: Tables $\k345$ -lb-tbl.sas



# Table 14.3.4.1 - Abnormal laboratory values - Safety set

**Category of Laboratory Parameters: HEMATOLOGY** 

| Subject<br>ID | Time<br>Point | Collection<br>Date/time | Parameter | Value and<br>Abnormality <sup>1</sup> | Normal Range or<br>Reference Value | Clinically<br>Significant? |
|---|---|---|---|---|---|---|
| S001/001 | Screening | ddMMMyyyy hh:mm | Leukocytes [10^9/L] | 10.02 [H] | 4.00 - 10.00 | N |
| S001/001 | End of Study | <br>ddMMMyyyy hh:mm | <br>Leukocytes [10^9/L] | <br>10.02 [H] | 4.00 - 10.00 | <br>N |
| | | ••• | <b></b> | ••• | ••• | ••• |

Note 1: H=Higher than upper normal limit, L=Lower than lower normal limit

Source: Listing 16.2.8.1 - Individual laboratory measurements

Program: Tables\k345-lb-tbl.sas



# Table 14.3.4.1 - Abnormal laboratory values - Safety set

**Category of Laboratory Parameters: COAGULATION** 

| Subject<br>ID | Time<br>Point | Collection<br>Date/time | Parameter | Value and Abnormality <sup>1</sup> | Normal Range or<br>Reference Value | Clinically<br>Significant? |
|---|---|---|---|---|---|---|
| S001/001 | Screening | ddMMMyyyy hh:mm | Prothrombin time [sec] | 9.00 [L] | 10.00 - 13.00 | N |

Note 1: H=Higher than upper normal limit, L=Lower than lower normal limit

Source: Listing 16.2.8.1 - Individual laboratory measurements

 $Program: Tables \verb|\k345-lb-tbl.sas|$ 



# Table 14.3.4.1 - Abnormal laboratory values - Safety set

**Category of Laboratory Parameters: URINE ANALYSIS** 

| Subject | Time | Collection | Parameter | Value and | Normal Range or | Clinically |
|---|---|---|---|---|---|---|
| ID | Point | Date/time | | Abnormality <sup>1</sup> | Reference Value | Significant? |
| S001/001 | Screening | ddMMMyyyy hh:mm | Urinary Hemoglobin | +++ [A] | Absent | N |
| S001/001 | | | | | | |
| | End of Study | ddMMMyyyy hh:mm | Urinary Hemoglobin | +++ [A] | Absent | N |

Note 1: A=Different from reference value

Source: Listing 16.2.8.1 - Individual laboratory measurements

Program: Tables\k345-lb-tbl.sas



Table 14.3.4.2 - Contingency tables of investigator's interpretation of laboratory test results - Safety set

| Time Point | Investigator's interpretation | Safety Set<br>N=XX |
|---|---|---|
| Screening | Normal Abnormal, Not Clinically Significant Abnormal, Clinically Significant | nn (xx.x)<br>nn (xx.x)<br>nn (xx.x) |
| End of Study | Normal Abnormal, Not Clinically Significant Abnormal, Clinically Significant | nn (xx.x)<br>nn (xx.x)<br>nn (xx.x) |

Note: The number and the proportion of subjects for each classification level are reported

The denominator for calculating the proportions is the number of subjects in the safety set

Source: Listing 16.2.8.2 - Investigator's interpretation of laboratory test results

Program: Tables\k345-lb-tbl.sas



Table 14.3.5.1 - Abnormal vital signs - Safety set

| Subject<br>ID | Time<br>Point | Assessment Date/Time | Parameter | Value and<br>Abnormality <sup>1</sup> | Normal Range | Clinically Significant? |
|---|---|---|---|---|---|---|
| S001/001 | Screening | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 | N |
| S001/001 | Visit 3 - Day 1 - Pre-dose | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 | N |
| ••• | | | <del></del> | | ••• | ••• |

Note 1: H=Higher than upper normal limit, L=Lower than lower normal limit

Source: Listing 16.2.9.1 - Vital signs and body weight

Program: Tables\k345-vs-tbl.sas



Table 14.3.5.2 - Descriptive statistics of vital signs and body weight at screening, day -1 and end of study - Safety set

| Parameter | Time Point | Statistics | Safety Set<br>N=XX |
|---|---|---|---|
| Systolic Blood Pressure [mmHg] | Screening | N | nn |
| Σ y στο του Ε του του Ε του του Ε του του Ε του του Ε του του Ε του του του Ε του του του Ε του του του του του Ε του | 2000 | Mean | XXX.X |
| | | SD | XXX.X |
| | | CV% | XXX.X |
| | | Min | XXX |
| | | Median | XXX.X |
| | | Max | xxx |
| Systolic Blood Pressure [mmHg] | Day -1 | N | nn |
| Systems Blood Fressure [mmrig] | Duy 1 | Mean | XXX.X |
| | | SD | XXX.X |
| | | CV% | XXX.X |
| | | Min | XXX |
| | | Median | XXX.X |
| | | Max | XXX |
| Systolic Blood Pressure [mmHg] | End of Study | N | nn |
| , | , | Mean | XXX.X |
| | | SD | XXX.X |
| | | CV% | XXX.X |
| | | Min | XXX |
| | | Median | XXX.X |
| | | Max | XXX |

Note: End of Study = Visit 6 - Day 4 - 72 hour post-dose or early termination visit for vital signs, final visit or early termination visit for body weight

Source: Listing 16.2.9.1 - Vital signs and body weight

Program: Tables\k345-vs-tbl.sas



Table 14.3.5.2 - Descriptive statistics of vital signs and body weight at screening, day -1 and end of study - Safety set

| Parameter | Time Point | Statistics | Safety Set<br>N=XX |
|---|---|---|---|
| Diastolic Blood Pressure [mmHg] | Screening | N | nn |
| 2100011 2100011 [ | S • · | Mean | XXX.X |
| | | SD | XXX.X |
| | | CV% | XXX.X |
| | | Min | XXX |
| | | Median | XXX.X |
| | | Max | xxx |
| Diastolic Blood Pressure [mmHg] | Day -1 | N | nn |
| | | Mean | XXX.X |
| | | SD | XXX.X |
| | | CV% | XXX.X |
| | | Min | XXX |
| | | Median | XXX.X |
| | | Max | XXX |
| Diagtalia Dland Programa [mmHa] | End of Study | N | |
| Diastolic Blood Pressure [mmHg] | End of Study | | nn |
| | | Mean | XXX.X |
| | | SD | XXX.X |
| | | CV% | XXX.X |
| | | Min | XXX |
| | | Median | XXX.X |
| | | Max | XXX |

Note: End of Study = Visit 6 - Day 4 - 72 hour post-dose or early termination visit for vital signs, final visit or early termination visit for body weight

Source: Listing 16.2.9.1 - Vital signs and body weight

Program: Tables\k345-vs-tbl.sas



Table 14.3.5.2 - Descriptive statistics of vital signs and body weight at screening, day -1 and end of study - Safety set

| Parameter | Time Point | Statistics | Safety Set<br>N=XX |
|---|---|---|---|
| Heart Rate [beats/min] | Screening | N | nn |
| 110010 11000 [0 0000 11111] | 5 <b>4.44</b> 5 | Mean | XXX.X |
| | | SD | XXX.X |
| | | CV% | XXX.X |
| | | Min | XXX |
| | | Median | XXX.X |
| | | Max | xxx |
| Heart Rate [beats/min] | Day -1 | N | nn |
| | | Mean | XXX.X |
| | | SD | XXX.X |
| | | CV% | XXX.X |
| | | Min | XXX |
| | | Median | XXX.X |
| | | Max | XXX |
| Heart Rate [beats/min] | End of Study | N | nn |
| Heart Rate [beats/film] | Elia of Study | | |
| | | Mean | XXX.X |
| | | SD | XXX.X |
| | | CV% | XXX.X |
| | | Min | XXX |
| | | Median | XXX.X |
| | | Max | XXX |

Note: End of Study = Visit 6 - Day 4 - 72 hour post-dose or early termination visit for vital signs, final visit or early termination visit for body weight

Source: Listing 16.2.9.1 - Vital signs and body weight

Program: Tables\k345-vs-tbl.sas



Table 14.3.5.2 - Descriptive statistics of vital signs and body weight at screening, day -1 and end of study - Safety set

| Parameter | Time Point | | Statistics | Safety Set<br>N=XX |
|-----------------|--------------|---------|------------|--------------------|
| Temperature [C] | Screening | | N | nn |
| remperature [e] | Sercening | | Mean | XXX.X |
| | | | SD | XXX.X |
| | | | CV% | XXX.X |
| | | | Min | XXX |
| | | | Median | XXX.X |
| | | | Max | XXX |
| Temperature [C] | Screening | < 37.5 | n (%) | nn (xx.x) |
| | - | >= 37.5 | n (%) | nn (xx.x) |
| Temperature [C] | Day -1 | | N | nn |
| | , | | Mean | XXX.X |
| | | | SD | XXX.X |
| | | | CV% | XXX.X |
| | | | Min | XXX |
| | | | Median | XXX.X |
| | | | Max | XXX |
| Temperature [C] | Day -1 | < 37.5 | n (%) | nn (xx.x) |
| | Ž | >= 37.5 | n (%) | nn (xx.x) |
| Temperature [C] | End of Study | | N | nn |

Note: End of Study = Visit 6 - Day 4 - 72 hour post-dose or early termination visit for vital signs, final visit or early termination visit for body weight

Source: Listing 16.2.9.1 - Vital signs and body weight

Program: Tables\k345-vs-tbl.sas



Table 14.3.5.2 - Descriptive statistics of vital signs and body weight at screening, day -1 and end of study - Safety set

| Parameter | Time Point | | Statistics | Safety Set<br>N=XX |
|-----------------|--------------|---------|------------|--------------------|
| Temperature [C] | End of Study | | Mean | XXX.X |
| | | | SD | XXX.X |
| | | | CV% | XXX.X |
| | | | Min | XXX |
| | | | Median | XXX.X |
| | | | Max | XXX |
| Temperature [C] | End of Study | < 37.5 | n (%) | nn (xx.x) |
| | | >= 37.5 | n (%) | nn (xx.x) |
| Weight [kg] | Screening | | N | nn |
| | | | Mean | XXX.X |
| | | | SD | XXX.X |
| | | | CV% | XXX.X |
| | | | Min | xxx |
| | | | Median | XXX.X |
| | | | Max | XXX |
| Weight [kg] | End of Study | | N | nn |
| | , | | Mean | XXX.X |
| | | | SD | XXX.X |
| | | | CV% | XXX.X |
| | | | Min | XXX |

Note: End of Study = Visit 6 - Day 4 - 72 hour post-dose or early termination visit for vital signs, final visit or early termination visit for body weight

Source: Listing 16.2.9.1 - Vital signs and body weight

Program: Tables\k345-vs-tbl.sas



Table 14.3.5.2 - Descriptive statistics of vital signs and body weight at screening, day -1 and end of study - Safety set

| Parameter | Time Point | Statistics | Safety Set<br>N=XX |
|-------------|--------------|------------|--------------------|
| Weight [kg] | End of Study | Median | XXX.X |
| | | Max | XXX |

Note: End of Study = Visit 6 - Day 4 - 72 hour post-dose or early termination visit for vital signs, final visit or early termination visit for body weight

Source: Listing 16.2.9.1 - Vital signs and body weight

Program: Tables\k345-vs-tbl.sas



Table 14.3.5.3 - Descriptive statistics of vital signs during the study - Safety set

| | | | Safe | ty Set |
|---|---|---|---|---|
| Parameter | Time Point | Statistics | Ladarixin<br>fed (T)<br>N=XX | Ladarixin<br>fasting (R)<br>N=XX |
| Systolic Blood Pressure [mmHg] | Day 1 - Pre-dose | N | nn | nn |
| Systone Blood Fressure [mining] | Day 1 The dose | Mean | XXX.X | XXX.X |
| | | SD | XXX.X | XXX.X |
| | | CV% | XXX.X | XXX.X |
| | | Min | XXX | XXX |
| | | Median | XXX.X | |
| | | Max | | XXX.X |
| | | Iviax | XXX | XXX |
| Systolic Blood Pressure [mmHg] | Day 4 - 72 hour post-dose | N | nn | nn |
| | | Mean | XXX.X | XXX.X |
| | | SD | XXX.X | XXX.X |
| | | CV% | XXX.X | XXX.X |
| | | Min | XXX | XXX |
| | | Median | XXX.X | XXX.X |
| | | Max | xxx | xxx |
| Diastolic Blood Pressure [mmHg] | Day 1 - Pre-dose | N | nn | nn |
| | | Mean | XXX.X | XXX.X |
| | | SD | XXX.X | XXX.X |
| | | CV% | XXX.X | XXX.X |
| | | Min | XXX | XXX |
| | | Median | XXX.X | XXX.X |
| | | Max | XXX | XXX |

Note: Subjects are summarised according to the product they actually received

Source: Listing 16.2.9.1 - Vital signs and body weight

Program: Tables\k345-vs-tbl.sas



Table 14.3.5.3 - Descriptive statistics of vital signs during the study - Safety set

| | | | Safe | ty Set |
|---|---|---|---|---|
| Parameter | Time Point | Statistics | Ladarixin<br>fed (T)<br>N=XX | Ladarixin<br>fasting (R)<br>N=XX |
| Diastolic Blood Pressure [mmHg] | Day 4 - 72 hour post-dose | N | nn | nn |
| [ | - mj · · · - seem prese meet | Mean | XXX.X | XXX.X |
| | | SD | XXX.X | XXX.X |
| | | CV% | XXX.X | XXX.X |
| | | Min | XXX | XXX |
| | | Median | XXX.X | XXX.X |
| | | Max | XXX | XXX |
| Heart Rate [beats/min] | Day 1 - Pre-dose | N | nn | nn |
| | <u>, </u> | Mean | XXX.X | XXX.X |
| | | SD | XXX.X | XXX.X |
| | | CV% | XXX.X | XXX.X |
| | | Min | XXX | XXX |
| | | Median | XXX.X | XXX.X |
| | | Max | XXX | XXX |
| Heart Rate [beats/min] | Day 4 - 72 hour post-dose | N | nn | nn |
| | 1 | Mean | XXX.X | XXX.X |
| | | SD | XXX.X | XXX.X |
| | | CV% | XXX.X | XXX.X |
| | | Min | XXX | XXX |
| | | Median | XXX.X | XXX.X |
| | | Max | XXX | XXX |

Note: Subjects are summarised according to the product they actually received

Source: Listing 16.2.9.1 - Vital signs and body weight

Program: Tables\k345-vs-tbl.sas



Table 14.3.5.3 - Descriptive statistics of vital signs during the study - Safety set

| | | | Safe | ety Set |
|---|---|---|---|---|
| Parameter | Time Point | Statistics | Ladarixin<br>fed (T)<br>N=XX | Ladarixin<br>fasting (R)<br>N=XX |
| Temperature [C] | Day 1 - Pre-dose | N | nn | nn |
| remperature [C] | Day 1 - 11e-dose | Mean | XXX.X | XXX.X |
| | | SD | XXX.X<br>XXX.X | XXX.X |
| | | CV% | XXX.X<br>XXX.X | XXX.X |
| | | Min | | |
| | | Median | XXX | XXX |
| | | | XXX.X | XXX.X |
| | | Max | XXX | XXX |
| Temperature [C] | Day 1 - Pre-dose | < 37.5 n (%) | nn (xx.x) | nn (xx.x) |
| | | >= 37.5 n (%) | nn(xx.x) | nn (xx.x) |
| Temperature [C] | Day 4 - 72 hour post-dose | N | nn | nn |
| 1 2 3 | 7 | Mean | XXX.X | XXX.X |
| | | SD | XXX.X | XXX.X |
| | | CV% | XXX.X | XXX.X |
| | | Min | XXX | XXX |
| | | Median | XXX.X | XXX.X |
| | | Max | XXX | xxx |
| Temperature [C] | Day 4 - 72 hour post-dose | < 37.5 n (%) | nn (xx.x) | nn (xx.x) |
| 1 | , | >= 37.5 n (%) | nn(xx.x) | nn (xx.x) |

Note: Subjects are summarised according to the product they actually received

Source: Listing 16.2.9.1 - Vital signs and body weight

Program: Tables\k345-vs-tbl.sas



Table 14.3.5.4 - Contingency tables of investigator's interpretation of ECG at screening, day -1 and end of study - Safety set

| Time Point | Investigator's interpretation | Safety Set<br>N=XX |
|---|---|---|
| Screening | Normal Abnormal, Not Clinically Significant | nn (xx.x) |
| | Abnormal, Clinically Significant | nn (xx.x)<br>nn (xx.x) |
| Day -1 | Normal Abnormal, Not Clinically Significant Abnormal, Clinically Significant | nn (xx.x)<br>nn (xx.x)<br>nn (xx.x) |
| End of Study | Normal Abnormal, Not Clinically Significant Abnormal, Clinically Significant | nn (xx.x)<br>nn (xx.x)<br>nn (xx.x) |

Note: End of Study = Visit 6 - Day 4 - 72 hour post-dose or early termination visit

The number and the proportion of subjects for each classification level are reported

The denominator for calculating the proportions is the number of subjects in the safety set

Source: Listing 16.2.9.2 - Investigator's interpretation of ECG

Program: Tables\k345-eg-tbl.sas



Table 14.3.5.5 - Contingency tables of investigator's interpretation of ECG during the study - Safety set

| | | Safety Set | |
|---|---|---|---|
| Time Point | Investigator's interpretation | Ladarixin fed (T)<br>N=XX | Ladarixin fasting (R)<br>N=XX |
| Day 1 - Pre-dose | Normal | nn (xx.x) | nn (xx.x) |
| | Abnormal, Not Clinically Significant | nn (xx.x) | nn (xx.x) |
| | Abnormal, Clinically Significant | nn (xx.x) | nn (xx.x) |
| Day 4 - 72 hour post-dose | Normal | nn (xx.x) | nn (xx.x) |
| | Abnormal, Not Clinically Significant | nn (xx.x) | nn (xx.x) |
| | Abnormal, Clinically Significant | nn (xx.x) | nn (xx.x) |

Note The number and the proportion of subjects for each classification level are reported

The denominator for calculating the proportions is the number of subjects in the safety set of each treatment group

Source: Listing 16.2.9.2 - Investigator's interpretation of ECG

 $Program: Tables \backslash k345\text{-}eg\text{-}tbl.sas$ 



Table 14.3.5.6 - Descriptive statistics of dose per body weight - Safety set

| Parameter | Sex | Statistics | Safety Set<br>N=XX |
|---|---|---|---|
| Dose per body weight [mg/kg] | Females | N | nn |
| 1 7 2 1 2 23 | | Mean | XXX.X |
| | | SD | XXX.X |
| | | CV% | XXX.X |
| | | Median | XXX.X |
| | | Min | XXX |
| | | Max | xxx |
| Dose per body weight [mg/kg] | Males | N | nn |
| Dose per body weight [ing/kg] | Maics | Mean | XXX.X |
| | | SD | XXX.X |
| | | CV% | XXX.X |
| | | Median | XXX.X |
| | | Min | XXX |
| | | Max | |
| | | IVIAA | XXX |
| Dose per body weight [mg/kg] | Females and males | N | nn |
| | | Mean | XXX.X |
| | | SD | XXX.X |
| | | CV% | XXX.X |
| | | Median | XXX.X |
| | | Min | XXX |
| | | Max | xxx |

Note: The dose per body weight was calculated using the screening body weight

Source: Listing 16.2.5.2 - Dose per body weight

Program: Tables\k345-ex-tbl.sas



Table 14.3.5.7 - Descriptive statistics of wash-out - Safety set

| Parameter | Statistics | Safety Set<br>N=XX |
|---|---|---|
| Wash-out between IMP administration of Period 1 and Period 2 [days] | N<br>Min<br>Max | nn<br>xxx<br>xxx |

Note: The wash-out is calculated as the difference in days between the dates of product administrations

Source: Listing 16.2.5.1 - Investigational medicinal products administration

Program: Tables\k345-ex-tbl.sas



#### Section 16.2 - Individual Subject Data Listings Shells

| Listing 16.2.1.1 - Discontinued subjects |
|--------------------------------------------------------------------------|
| Listing 16.2.2.1 - Protocol deviations |
| Listing 16.2.2.2 - Assigned and actual sequence of treatments mismatches |
| Listing 16.2.3.1 - Subjects excluded from PK and/or safety analysis |
| Listing 16.2.4.1 - Subjects' disposition |
| Listing 16.2.4.2 - Analysis sets |
| Listing 16.2.4.3 - Demography |
| Listing 16.2.4.4 - Inclusion/Exclusion criteria not met |
| Listing 16.2.5.1 - Investigational medicinal products administration |
| Listing 16.2.5.2 - Dose per body weight |
| Listing 16.2.5.3 - PK samples collection dates and times |

Listing 16.2.5.4 - Total DF 2156Y concentrations (µg/mL) measured in plasma

Listing 16.2.5.5 - Unbound DF 2156Y concentrations (µg/mL) measured in plasma

Listing 16.2.5.6 - DF 2108Y concentrations ( $\mu g/mL$ ) measured in plasma

Listing 16.2.5.7 - DF 2227Y concentrations (µg/mL) measured in plasma

Listing 16.2.6.1 - Total DF 2156Y plasma PK parameters

Listing 16.2.6.2 - DF 2108Y plasma PK parameters

Listing 16.2.6.3 - DF 2227Y plasma PK parameters

Listing 16.2.6.4 - Total DF 2156Y, DF 2108Y and DF 2227Y relative bioavailability in plasma calculated as AUC0-t T/R ratio

Listing 16.2.7.1 - Treatment-emergent adverse events

Listing 16.2.7.2 - Pre-treatment adverse events

Listing 16.2.8.1 - Individual laboratory measurements

Listing 16.2.8.2 - Investigator's interpretation of laboratory test results

Listing 16.2.9.1 - Vital signs and body weight

Listing 16.2.9.2 - Investigator's interpretation of ECG

Listing 16.2.9.3 - Abnormal ECG parameters

Listing 16.2.10.1 - Medical and surgical history

Listing 16.2.10.2 - Physical examination

Listing 16.2.10.3 - Prior and concomitant medications

Listing 16.2.10.4 - Subjects study visits


Statistical analysis plan CRO-PK-20-345 Sponsor code LDX0219 Ladarixin 200 mg capsules - food effect Final version 1.0, 10FEB21



Section 16.2 - Individual Subject Data Listings Shells

Listing 16.2.10.5 - Fertility status and contraception Listing 16.2.10.6 - Meals



**Listing 16.2.1.1 - Discontinued subjects** 

| Subject<br>ID | Last IMP before discontinuation | Sex | Age<br>(years) | Last<br>visit | Time elapsed from last drug administration | Date of premature | Primary reason for subject premature study termination |
|---|---|---|---|---|---|---|---|
| | | | | | (days) | discontinuation | |
| S001/001 | Ladarixin fed (T) | M | 30 | Visit 3 | 1 | ddMMMyyyy | Withdrawal by subject |
| S003/002 | Ladarixin fasting (R) | F | 27 | Visit 5 | 2 | ddMMMyyyy | Adverse event |
| S005/004 | Ladarixin fasting (R) | M | 18 | Visit 3 | 2 | ddMMMyyyy | Physician decision |
| S007/006 | Ladarixin fed (T) | F | 27 | Visit 5 | 2 | ddMMMyyyy | Adverse event |
| S011/010 | Ladarixin fasting (R) | M | 18 | Visit 3 | 2 | ddMMMyyyy | Physician decision |
| | | ••• | | ••• | | ••• | |

Note: Subjects are listed according to the last product they actually received before discontinuation

Program: Listings\k345-ds-lst.sas



**Listing 16.2.2.1 - Protocol deviations** 

| Subject<br>ID | Deviation<br>Number | Deviation<br>Category | Deviation<br>Coded<br>Term | Deviation Description |
|---|---|---|---|---|
| S001/001 | 1 | Minor | Deviation from scheduled sampling time | Sample number 2 was collected outside the window of 15 min post-dose |
| S007/006 | 1 | Major | Inclusion criteria violation | Inclusion criteria violation |

Program: Listings\k345-dv-lst.sas



# Listing 16.2.2.2 - Assigned and actual sequence of treatments mismatches

| Subject<br>ID | Assigned Sequence of Treatments | Actual Sequence of Treatments |
|---|---|---|
| S003/002 | Ladarixin fed (T) - Ladarixin fasting (R) | Ladarixin fasting (R) - Ladarixin fed (T) |
| | <del></del> | |

Program: Listings\k345-ds-lst.sas



Listing 16.2.3.1 - Subjects excluded from PK and/or safety analysis

| Subject<br>ID | Sex | Age<br>(years) | Enrolled<br>Set | Safety<br>Set | PK<br>Set 1 | PK<br>Set 2 | Reason for the exclusion |
|---|---|---|---|---|---|---|---|
| S010/008 | F | 30 | Y | N | N | N | Lack of IMP administration |
| S015/013 | F | 20 | Y | Y | Y | Y | Major protocol deviations |
| | ••• | | • | • | • | | |

Program: Listings\k345-ds-lst.sas



# Listing 16.2.4.1 - Subjects' disposition

| Subject<br>ID | Date of<br>Informed | Date of Screening | Date of<br>Enrolment | Date of<br>First | Date of<br>Last | Completed or | Date of Study<br>Completion or | Date of<br>End of | Reason for discontinuation |
|---|---|---|---|---|---|---|---|---|---|
| | Consent | | | Administration | Administration | Discontinued | Discontinuation | Participation | |
| S001/001 | ddMMMyyyy | ddMMMyyyy | ddMMMyyyy | ddMMMyyyy | ddMMMyyyy | Discontinued | ddMMMyyyy | ddMMMyyyy | Withdrawal by subject |
| S002/002 | ddMMMyyyy | ddMMMyyyy | ddMMMyyyy | ddMMMyyyy | ddMMMyyyy | Completed | ddMMMyyyy | ddMMMyyyy | |
| S005/003 | ddMMMyyyy | ddMMMyyyy | ddMMMyyyy | ddMMMyyyy | ddMMMyyyy | Discontinued | ddMMMyyyy | ddMMMyyyy | Adverse event |

Program: Listings\k345-ds-lst.sas



# Listing 16.2.4.2 - Analysis sets

| Subject | Planned Sequence | Enrolled | Safety | PK | PK | Reason for the exclusion |
|---|---|---|---|---|---|---|
| ID | | Set | Set | Set 1 | Set 2 | |
| S001/001 | Ladarixin fed (T) - Ladarixin fasting (R) | Y | N | N | N | Lack of IMP intake |
| S003/002 | Ladarixin fasting (R) - Ladarixin fed (T) | Y | Y | Y | Y | |
| ••• | | • | • | | • | |

Note: Subjects are listed according to the sequence they were assigned to

Program: Listings\k345-ds-lst.sas



# Listing 16.2.4.3 - Demography

| Subject<br>ID | Sex | Race | Birth<br>Year | Age<br>(years) | Height (cm) | Body Weight (kg) | Body Mass Index (kg/m²) |
|---|---|---|---|---|---|---|---|
| S001/001 | F | White | 2001 | 19 | 170 | 55.0 | 19.0 |
| S002/002 | M | White | 1990 | 30 | 187 | 91.0 | 26.0 |

Note:Program:Listings\k345-dm-lst.sas



# Listing 16.2.4.4 - Inclusion/Exclusion criteria not met

| Subject<br>ID | Criterion | Verbatim |
|---|---|---|
| S001/001 | Inclusion criterion 3 | Body Mass Index (BMI): 18.5-30 kg/m2 inclusive |
| | ••• | <del></del> |

Program: Listings\k345-ie-lst.sas



# Listing 16.2.5.1 - Investigational medicinal products administration

**Investigational Medicinal Product: Ladarixin fed (T)** 

| Subject<br>ID | Adm.<br>Nr. | Administration<br>Time Point | Administration<br>Date/time | Breakfast<br>Start<br>Date/time | Time from<br>Start of<br>Breakfast | Fasting Conditions<br>Start Date/time | Time from<br>Start of<br>Fasting<br>Conditions | Fasting Conditions<br>From 10 h before<br>IMP<br>Administration? |
|---|---|---|---|---|---|---|---|---|
| S001/001 | 1 | Visit 3 - Day 1 - $08:00 \pm 1$ hour | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | xx min | | | |
| ••• | ••• | ··· | ••• | ••• | ••• | ••• | ••• | ••• |

Note: Subjects are listed according to the product they actually received

Program: Listings\k345-ex-lst.sas


## Listing 16.2.5.1 - Investigational medicinal products administration

**Investigational Medicinal Product: Ladarixin fasting (R)** 

| Subject<br>ID | Adm.<br>Nr. | Administration<br>Time Point | Administration<br>Date/time | Breakfast<br>Start<br>Date/time | Time from<br>Start of<br>Breakfast | Fasting Conditions<br>Start Date/time | Time from<br>Start of<br>Fasting<br>Conditions | Fasting Conditions From 10 h before IMP Administration? |
|---|---|---|---|---|---|---|---|---|
| S001/001 | 2 | Visit 6 - Day 1 - $08:00 \pm 1$ hour | ddMMMyyyy hh:mm | | | ddMMMyyyy hh:mm | xx h xx min | Y |
| ••• | ••• | | ••• | ••• | ••• | ••• | ••• | ••• |

Note: Subjects are listed according to the product they actually received

Program: Listings\k345-ex-lst.sas



## Listing 16.2.5.2 - Dose per body weight

| Subject<br>ID | Active<br>Ingredient | Dose<br>Administered | Body Weight at Screening | Dose per<br>Body Weight |
|---|---|---|---|---|
| | _ | (mg) | (kg) | (mg/kg) |
| S001/001 | Ladarixin | 800 | 55.0 | 14.54 |

Note: The dose per body weight is calculated using the screening body weight

Program: Listings\k345-ex-lst.sas



Listing 16.2.5.3 - PK samples collection dates and times

**Investigational Medicinal Product: Ladarixin fed (T)** 

| Subject<br>ID | IMP Administration<br>Date/Time | IMP Adm<br>Nr. | Time Point | Sample<br>Number | Collection<br>Date/time | Time from IMP Administration |
|---|---|---|---|---|---|---|
| S001/001 | ddMMMyyyy hh:mm | 1 | Pre-dose - Within 30 min before IMP administration | 1 | ddMMMyyyy hh:mm | -xx min |
| S001/001 | ddMMMyyyy hh:mm | 1 | 15 min post-dose | 2 | ddMMMyyyy hh:mm | xx min |
| S001/001 | ddMMMyyyy hh:mm | 1 | 30 min post-dose $\pm 1$ min | 3 | ddMMMyyyy hh:mm | xx min |
| S001/001 | ddMMMyyyy hh:mm | 1 | 1 hour post-dose $\pm$ 3 min | 4 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 1 | 1.5 hour post-dose $\pm$ 3 min | 5 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 1 | 2 hours post-dose $\pm$ 5 min | 6 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 1 | 3 hours post-dose $\pm$ 5 min | 7 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 1 | 4 hours post-dose $\pm$ 5 min | 8 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 1 | 5 hours post-dose $\pm$ 5 min | 9 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 1 | 6 hours post-dose $\pm$ 5 min | 10 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 1 | 8 hours post-dose $\pm$ 10 min | 11 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 1 | 10 hours post-dose $\pm$ 10 min | 12 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 1 | 12 hours post-dose $\pm$ 10 min | 13 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 1 | 18 hours post-dose $\pm$ 10 min | 14 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 1 | 24 hours post-dose $\pm$ 10 min | 15 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 1 | 30 hours post-dose $\pm$ 10 min | 16 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 1 | $36 \text{ min post-dose} \pm 30 \text{ min}$ | 17 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 1 | 48 hour post-dose $\pm$ 30 min | 18 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 1 | 54 hour post-dose $\pm$ 30 min | 19 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 1 | 60 hours post-dose $\pm$ 30 min | 20 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 1 | 72 hours post-dose $\pm$ 30 min | 21 | ddMMMyyyy hh:mm | xx h xx min |
| | | | | | | ••• |

Note: Subjects are listed according to the product they actually received

Program: Listings\k345-pc-lst.sas



Listing 16.2.5.3 - PK samples collection dates and times

**Investigational Medicinal Product: Ladarixin fasting (R)** 

| Subject<br>ID | IMP Administration<br>Date/Time | IMP Adm<br>Nr. | Time Point | Sample<br>Number | Collection Date/time | Time from IMP Administration |
|---|---|---|---|---|---|---|
| S001/001 | ddMMMyyyy hh:mm | 2 | Pre-dose - Within 30 min before IMP administration | 22 | ddMMMyyyy hh:mm | -xx min |
| S001/001 | ddMMMyyyy hh:mm | 2 | 15 min post-dose | 23 | ddMMMyyyy hh:mm | xx min |
| S001/001 | ddMMMyyyy hh:mm | 2 | 30 min post-dose $\pm 1$ min | 24 | ddMMMyyyy hh:mm | xx min |
| S001/001 | ddMMMyyyy hh:mm | 2 | 1 hour post-dose $\pm$ 3 min | 25 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 2 | 1.5 hour post-dose $\pm$ 3 min | 26 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 2 | 2 hours post-dose $\pm$ 5 min | 27 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 2 | 3 hours post-dose $\pm$ 5 min | 28 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 2 | 4 hours post-dose $\pm$ 5 min | 29 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 2 | 5 hours post-dose $\pm$ 5 min | 30 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 2 | 6 hours post-dose $\pm$ 5 min | 31 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 2 | 8 hours post-dose $\pm$ 10 min | 32 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 2 | 10 hours post-dose $\pm$ 10 min | 33 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 2 | 12 hours post-dose $\pm$ 10 min | 34 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 2 | 18 hours post-dose $\pm$ 10 min | 35 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 2 | 24 hours post-dose $\pm$ 10 min | 36 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 2 | 30 hours post-dose $\pm$ 10 min | 37 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 2 | $36 \text{ min post-dose} \pm 30 \text{ min}$ | 38 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 2 | 48 hour post-dose $\pm$ 30 min | 39 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 2 | $54 \text{ hour post-dose} \pm 30 \text{ min}$ | 40 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 2 | 60 hours post-dose $\pm$ 30 min | 41 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 2 | 72 hours post-dose $\pm$ 30 min | 42 | ddMMMyyyy hh:mm | xx h xx min |
| ••• | | | | | ••• | ••• |

Note: Subjects are listed according to the product they actually received

Program: Listings\k345-pc-lst.sas



## Listing 16.2.5.4 - Total DF 2156Y concentrations (µg/mL) measured in plasma

**Investigational Medicinal Product: Ladarixin fed (T)** 

| Subject<br>ID | Period | Pre<br>dose | 0.25 h | 0.5 h | 1 h | 1.5 h | 2 h | 3 h | 4 h | 5 h | 6 h | 8 h | 10 h | 12 h | 18 h | 24 h | 30 h | 36 h | 48 h | 54 h | 60 h | 72 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| S001/001 | 1 | BLQL | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | | | | | | ••• | | | | | | | | | | | | | | | | ••• |

BLQL: Below Lower Quantification Limit (x.xx µg/mL)

Program: pk-analysis\k345-tlf.sas



## Listing 16.2.5.4 - Total DF 2156Y concentrations (µg/mL) measured in plasma

**Investigational Medicinal Product: Ladarixin fasting (R)** 

| Subject<br>ID | Period | Pre<br>dose | 0.25 h | 0.5 h | 1 h | 1.5 h | 2 h | 3 h | 4 h | 5 h | 6 h | 8 h | 10 h | 12 h | 18 h | 24 h | 30 h | 36 h | 48 h | 54 h | 60 h | 72 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| S001/001 | 2 | BLQL | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| ••• | | ••• | | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• |

BLQL: Below Lower Quantification Limit (x.xx µg/mL)

Program: pk-analysis\k345-tlf.sas



# Listing 16.2.5.5 - Unbound DF 2156Y concentrations (µg/mL) measured in plasma

**Investigational Medicinal Product: Ladarixin fed (T)** 

| Subject Period<br>ID | 1 h | 3 h | 6 h | 12 h | 24 h |
|----------------------|-------|-------|-------|-------|-------|
| S001/001 1 | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |

BLQL: Below Lower Quantification Limit (x.xx µg/mL)

Program: pk-analysis\k345-tlf.sas



# Listing 16.2.5.5 - Unbound DF 2156Y concentrations (µg/mL) measured in plasma

**Investigational Medicinal Product: Ladarixin fasting (R)** 

| Subject Period<br>ID | 1 h | 3 h | 6 h | 12 h | 24 h |
|----------------------|-------|-------|-------|-------|-------|
| S001/001 2 | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |

BLQL: Below Lower Quantification Limit (x.xx µg/mL)

Program: pk-analysis\k345-tlf.sas



## Listing 16.2.5.6 - DF 2108Y concentrations (µg/mL) measured in plasma

**Investigational Medicinal Product: Ladarixin fed (T)** 

| Subject<br>ID | Period | Pre<br>dose | 0.25 h | 0.5 h | 1 h | 1.5 h | 2 h | 3 h | 4 h | 5 h | 6 h | 8 h | 10 h | 12 h | 18 h | 24 h | 30 h | 36 h | 48 h | 54 h | 60 h | 72 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| S001/001 | 1 | BLQL | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | | | | | | ••• | | | | | | | | | | | | | | | | ••• |

BLQL: Below Lower Quantification Limit (x.xx µg/mL)

Program: pk-analysis\k345-tlf.sas



## Listing 16.2.5.6 - DF 2108Y concentrations (µg/mL) measured in plasma

**Investigational Medicinal Product: Ladarixin fasting (R)** 

| Subject<br>ID | Period | Pre<br>dose | 0.25 h | 0.5 h | 1 h | 1.5 h | 2 h | 3 h | 4 h | 5 h | 6 h | 8 h | 10 h | 12 h | 18 h | 24 h | 30 h | 36 h | 48 h | 54 h | 60 h | 72 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| S001/001 | 2 | BLQL | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | | | | | | ••• | | | | | | | | | | | | | | | | ••• |

BLQL: Below Lower Quantification Limit (x.xx µg/mL)

Program: pk-analysis\k345-tlf.sas



## Listing 16.2.5.7 - DF 2227Y concentrations (µg/mL) measured in plasma

**Investigational Medicinal Product: Ladarixin fed (T)** 

| Subject<br>ID | Period | Pre<br>dose | 0.25 h | 0.5 h | 1 h | 1.5 h | 2 h | 3 h | 4 h | 5 h | 6 h | 8 h | 10 h | 12 h | 18 h | 24 h | 30 h | 36 h | 48 h | 54 h | 60 h | 72 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| S001/001 | 1 | BLQL | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| ••• | | ••• | | ••• | ••• | ••• | | ••• | ••• | ••• | ••• | ••• | | | ••• | | ••• | ••• | ••• | ••• | ••• | ••• |

BLQL: Below Lower Quantification Limit (x.xx µg/mL)

Program: pk-analysis\k345-tlf.sas



## Listing 16.2.5.7 - DF 2227Y concentrations (µg/mL) measured in plasma

**Investigational Medicinal Product: Ladarixin fasting (R)** 

| Subject<br>ID | Period | Pre<br>dose | 0.25 h | 0.5 h | 1 h | 1.5 h | 2 h | 3 h | 4 h | 5 h | 6 h | 8 h | 10 h | 12 h | 18 h | 24 h | 30 h | 36 h | 48 h | 54 h | 60 h | 72 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| S001/001 | 2 | BLQL | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | | | | | | ••• | | | | | | | | | | | | | | | | ••• |

BLQL: Below Lower Quantification Limit (x.xx µg/mL)

Program: pk-analysis\k345-tlf.sas



#### Listing 16.2.6.1 - Total DF 2156Y plasma PK parameters

## Investigational Medicinal Product: Ladarixin fed (T)

| Subject<br>ID | C <sub>max</sub><br>(μg/mL) | t <sub>max</sub><br>(h) | AUC <sub>0-t</sub><br>(h*μg/mL) | AUC <sub>0-inf</sub><br>(h*μg/mL) | AUCextra<br>(%) | t½<br>(h) | • z<br>(1/h) | Points | $\mathbb{R}^2$ |
|---|---|---|---|---|---|---|---|---|---|
| S001/001 | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| | | | | | | | ••• | | |

Note: Only subjects included in PK Set 1 are listed

Program: pk-analysis\k345-tlf.sas



#### Listing 16.2.6.1 - Total DF 2156Y plasma PK parameters

## Investigational Medicinal Product: Ladarixin fasting (R)

| Subject<br>ID | C <sub>max</sub><br>(μg/mL) | t <sub>max</sub><br>(h) | AUC <sub>0-t</sub><br>(h*μg/mL) | AUC <sub>0-inf</sub><br>(h*μg/mL) | AUCextra<br>(%) | t½<br>(h) | • z<br>(1/h) | Points | $\mathbb{R}^2$ |
|---|---|---|---|---|---|---|---|---|---|
| S001/001 | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| | | | | | | | ••• | | |

Note: Only subjects included in PK Set 1 are listed

Program: pk-analysis\k345-tlf.sas



## Listing 16.2.6.2 - DF 2108Y plasma PK parameters

## Investigational Medicinal Product: Ladarixin fed (T)

| Subject<br>ID | C <sub>max</sub><br>(µg/mL) | t <sub>max</sub><br>(h) | AUC <sub>0-t</sub><br>(h*µg/mL) | AUC <sub>0-inf</sub><br>(h*μg/mL) | AUCextra<br>(%) | t½<br>(h) | · <sub>z</sub> (1/h) | Points | $\mathbb{R}^2$ |
|---|---|---|---|---|---|---|---|---|---|
| S001/001 | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |

Note: Only subjects included in PK Set 2 are listed

Program: pk-analysis\k345-tlf.sas



## Listing 16.2.6.2 - DF 2108Y plasma PK parameters

## Investigational Medicinal Product: Ladarixin fasting (R)

| Subject<br>ID | C <sub>max</sub><br>(µg/mL) | t <sub>max</sub><br>(h) | AUC <sub>0-t</sub><br>(h*µg/mL) | AUC <sub>0-inf</sub><br>(h*μg/mL) | AUCextra<br>(%) | t½<br>(h) | · <sub>z</sub> (1/h) | Points | $\mathbb{R}^2$ |
|---|---|---|---|---|---|---|---|---|---|
| S001/001 | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |

Note: Only subjects included in PK Set 2 are listed

Program: pk-analysis\k345-tlf.sas



## Listing 16.2.6.3 - DF 2227Y plasma PK parameters

## Investigational Medicinal Product: Ladarixin fed (T)

| Subject<br>ID | C <sub>max</sub><br>(μg/mL) | t <sub>max</sub><br>(h) | AUC <sub>0-t</sub><br>(h*μg/mL) | AUC <sub>0-inf</sub><br>(h*μg/mL) | AUCextra<br>(%) | t½<br>(h) | • z<br>(1/h) | Points | R <sup>2</sup> |
|---|---|---|---|---|---|---|---|---|---|
| S001/001 | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| ••• | | ••• | | | | | | | |

Note: Only subjects included in PK Set 2 are listed

Program: pk-analysis\k345-tlf.sas



## Listing 16.2.6.3 - DF 2227Y plasma PK parameters

## Investigational Medicinal Product: Ladarixin fasting (R)

| Subject<br>ID | C <sub>max</sub><br>(μg/mL) | t <sub>max</sub><br>(h) | AUC <sub>0-t</sub><br>(h*μg/mL) | AUC <sub>0-inf</sub><br>(h*μg/mL) | AUCextra<br>(%) | t½<br>(h) | • z<br>(1/h) | Points | $\mathbb{R}^2$ |
|---|---|---|---|---|---|---|---|---|---|
| S001/001 | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| | | | | | | | ••• | | |

Note: Only subjects included in PK Set 2 are listed

Program: pk-analysis\k345-tlf.sas



#### Listing 16.2.6.4 - Total DF 2156Y, DF 2108Y and DF 2227Y relative bioavailability in plasma calculated as AUC<sub>0-t</sub> T/R ratio

| Subject ID | DF 2156Y Fred<br>(%) | DF 2108Y Fred (%) | DF 2227Y Fred (%) |
|------------|----------------------|-------------------|-------------------|
| S001/001 | XXX.XX | XXX.XX | XXX.XX |
| | ··· | | |

T: Ladarixin fed (T)

R: Ladarixin fasting (R)

Program: pk-analysis\k345-tlf.sas



## Listing 16.2.7.1 - Treatment-emergent adverse events

**Investigational Product: Ladarixin fed (T)** 

| Subject<br>ID | Adverse<br>Event<br>ID | | |
|---|---|---|---|
| S001/001 | 1 | Description: | Headache |
| | | AE Record date and time: | ddMMMyyyy hh:mm |
| | | Body Location: | Head |
| | | Preferred Term <sup>1</sup> : | Headache |
| | | System Organ Class <sup>1</sup> : | Nervous system disorders |
| | | Serious? | N |
| | | Frequency: | Continuous |
| | | Severity: | Mild |
| | | Action taken with Study Drug: | Dose not changed |
| | | Relationship with Investigational Study Drug? | Unlikely (remote) |
| | | Corrective therapy? | Y |
| | | Other Action Taken: | |
| | | Outcome: | Resolved |
| | | Start - End Date/Time (Day): | ddMMMyyyy hh:mm (k) - ddMMMyyyy hh:mm (k+n) |
| | | Did this Adverse Event result in discontinuation of the subject from the study? | N |

Note: Subjects are listed according to the product they actually received

Note 1: MedDRA version 23.1 Program: Listings\k345-ae-lst.sas



## Listing 16.2.7.1 - Treatment-emergent adverse events

## **Investigational Product: Ladarixin fasting (R)**

| Subject<br>ID | Adverse<br>Event<br>ID | | |
|---|---|---|---|
| S001/001 | 2 | Description: | Headache |
| | | AE Record date and time: | ddMMMyyyy hh:mm |
| | | Body Location: | Head |
| | | Preferred Term <sup>1</sup> : | Headache |
| | | System Organ Class <sup>1</sup> : | Nervous system disorders |
| | | Serious? | N |
| | | Frequency: | Continuous |
| | | Severity: | Mild |
| | | Action taken with Study Drug: | Dose not changed |
| | | Relationship with Investigational Study Drug? | Unlikely (remote) |
| | | Corrective therapy? | Y |
| | | Other Action Taken: | |
| | | Outcome: | Resolved |
| | | Start - End Date/Time (Day): | ddMMMyyyy hh:mm (k) - ddMMMyyyy hh:mm (k+n) |
| | | Did this Adverse Event result in discontinuation of the subject from the study? | N |

Note: Subjects are listed according to the product they actually received

Note 1: MedDRA version 23.1 Program: Listings\k345-ae-lst.sas



## Listing 16.2.7.2 - Pre-treatment adverse events

| Subject<br>ID | Adverse<br>Event<br>ID | | |
|---|---|---|---|
| S001/001 | 1 | Description: | Headache |
| | | AE Record date and time: | ddMMMyyyy hh:mm |
| | | Body Location: | Head |
| | | Preferred Term <sup>1</sup> : | Headache |
| | | System Organ Class <sup>1</sup> : | Nervous system disorders |
| | | Serious? | N |
| | | Frequency: | Continuous |
| | | Severity: | Mild |
| | | Action taken with Study Drug: | Dose not changed |
| | | Relationship with Investigational Study Drug? | Unlikely (remote) |
| | | Corrective therapy? | Y |
| | | Other Action Taken: | |
| | | Outcome: | Resolved |
| | | Start - End Date/Time (Day): | ddMMMyyyy hh:mm (k) - ddMMMyyyy hh:mm (k+n) |
| | | Did this Adverse Event result in discontinuation of the subject from the study? | N |

Note 1: MedDRA version 23.1 Program: Listings\k345-ae-lst.sas



**Listing 16.2.8.1 - Individual laboratory measurements** 

Category of Laboratory Parameters: BLOOD CHEMISTRY

| Subject<br>ID | Time<br>Point | Collection<br>Date/time | Parameter | Value and<br>Abnormality <sup>1</sup> | Normal Range or<br>Reference Value | Clinically<br>Significant? |
|---|---|---|---|---|---|---|
| S001/001 | Screening | ddMMMyyyy hh:mm | Sodium [mmol/L] | 138 [N] | 136 - 145 | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Potassium [mmol/L] | 4.4 [N] | 3.5 - 5.1 | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Calcium [mmol/L] | 2.27 [N] | 2.10 - 2.55 | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Chloride [mmol/L] | 103 [N] | 96 - 110 | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Phosphate [mmol/L] | 0.84 [L] | 0.87 - 1.45 | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Alkaline Phosphatase [U/L] | 95 [N] | <= 129 | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Gamma Glutamyl Transferase [U/L] | 17 [N] | <= 66 | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Aspartate Aminotransferase [U/L] | 24 [N] | <= 50 | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Alanine Aminotransferase [U/L] | 30 [N] | <= 50 | N |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Sodium [mmol/L] | 138 [N] | 136 - 145 | N |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Potassium [mmol/L] | 4.4 [N] | 3.5 - 5.1 | N |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Calcium [mmol/L] | 2.27 [N] | 2.10 - 2.55 | N |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Chloride [mmol/L] | 103 [N] | 96 - 110 | N |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Phosphate [mmol/L] | 0.84 [L] | 0.87 - 1.45 | N |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Alkaline Phosphatase [U/L] | 95 [N] | <= 129 | N |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Gamma Glutamyl Transferase [U/L] | 17 [N] | <= 66 | N |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Aspartate Aminotransferase [U/L] | 24 [N] | <= 50 | N |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Alanine Aminotransferase [U/L] | 30 [N] | <= 50 | N |

Note 1: N=Normal, H=Higher than upper normal limit, L=Lower than lower normal limit

 $Program: Listings \verb|\k345-lb-lst.sas|$ 



**Listing 16.2.8.1 - Individual laboratory measurements** 

Category of Laboratory Parameters: HEMATOLOGY

| Subject<br>ID | Time<br>Point | Collection<br>Date/time | Parameter | Value and<br>Abnormality <sup>1</sup> | Normal Range or<br>Reference Value | Clinically<br>Significant? |
|---|---|---|---|---|---|---|
| S001/001 | Screening | ddMMMyyyy hh:mm | Leukocytes [10^9/L] | 10.02 [H] | 4.00 - 10.00 | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Erythrocytes [10^12/L] | 5.19 [N] | 4.30 - 5.90 | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Hemoglobin [g/dL] | 15.4 [N] | 14.0 - 18.0 | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Hemoglobin [mmol/L] | 9.6 [N] | 8.7 - 11.2 | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Hematocrit [%] | 44 [N] | 42 - 52 | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Ery. Mean Corpuscular Volume [fL] | 84 [N] | 83 - 100 | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Ery. Mean Corpuscular Hemoglobin [pg] | 30 [N] | 27 - 34 | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Ery. Mean Corpuscular HGB Concentration [g/dL] | 35 [N] | 32 - 36 | N |
| | | | <del></del> | | | |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Leukocytes [10^9/L] | 10.02 [H] | 4.00 - 10.00 | N |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Erythrocytes [10 <sup>12</sup> /L] | 5.19 [N] | 4.30 - 5.90 | N |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Hemoglobin [g/dL] | 15.4 [N] | 14.0 - 18.0 | N |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Hemoglobin [mmol/L] | 9.6 [N] | 8.7 - 11.2 | N |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Hematocrit [%] | 44 [N] | 42 - 52 | N |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Ery. Mean Corpuscular Volume [fL] | 84 [N] | 83 - 100 | N |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Ery. Mean Corpuscular Hemoglobin [pg] | 30 [N] | 27 - 34 | N |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Ery. Mean Corpuscular HGB Concentration [g/dL] | 35 [N] | 32 - 36 | N |

Note 1: N=Normal, H=Higher than upper normal limit, L=Lower than lower normal limit

Program: Listings\k345-lb-lst.sas



#### **Listing 16.2.8.1 - Individual laboratory measurements**

**Category of Laboratory Parameters: COAGULATION** 

| Subject<br>ID | Time<br>Point | Collection<br>Date/time | Parameter | Value and <b>Abnormality</b> <sup>1</sup> | Normal Range or<br>Reference Value | Clinically Significant? |
|---|---|---|---|---|---|---|
| S001/001 | Screening | ddMMMyyyy hh:mm | Prothrombin time [sec] | 12.00 [N] | 10.00 - 13.00 | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | aPTT [sec] | 31.00 [N] | 30.00 - 40.00 | N |
| ••• | | | <b></b> | ••• | | ••• |

Note 1: N=Normal, H=Higher than upper normal limit, L=Lower than lower normal limit

Program: Listings\k345-lb-lst.sas



#### **Listing 16.2.8.1 - Individual laboratory measurements**

**Category of Laboratory Parameters: URINE ANALYSIS** 

| Subject<br>ID | Time<br>Point | Collection<br>Date/time | Parameter | Value and<br>Abnormality <sup>1</sup> | Normal Range or<br>Reference Value | Clinically<br>Significant? |
|---|---|---|---|---|---|---|
| S001/001 | Screening | ddMMMyyyy hh:mm | Urobilinogen | Normal [N] | Normal | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Urinary Bilirubin | Absent [N] | Absent | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Ketones | Absent [N] | Absent | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Urinary Hemoglobin | +++ [A] | Absent | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Urinary Leukocytes | Absent [N] | Absent | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Sediment Examination | Checked | | |
| S001/001 | Screening | ddMMMyyyy hh:mm | Urinary Sediment Leukocytes | Absent [N] | Absent or 0-2 per field | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Urinary Sediment Erythrocytes | 0-2 per field [N] | Absent or 0-2 per field | N |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Urobilinogen | Normal [N] | Normal | N |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Urinary Bilirubin | Absent [N] | Absent | N |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Ketones | Absent [N] | Absent | N |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Urinary Hemoglobin | +++ [A] | Absent | N |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Urinary Leukocytes | Absent [N] | Absent | N |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Sediment Examination | Checked | | |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Urinary Sediment Leukocytes | Absent [N] | Absent or 0-2 per field | N |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Urinary Sediment Erythrocytes | 0-2 per field [N] | Absent or 0-2 per field | N |

Note 1: N=Normal, A=Different from reference value

Program: Listings\k345-lb-lst.sas



#### Listing 16.2.8.1 - Individual laboratory measurements

Category of Laboratory Parameters: URINE DRUG SCREENING

| Subject<br>ID | Time<br>Point | Collection<br>Date/time | Parameter | Value and<br>Abnormality <sup>1</sup> | Normal Range or<br>Reference Value | Clinically<br>Significant? |
|---|---|---|---|---|---|---|
| S001/001 | Screening | ddMMMyyyy hh:mm | Amphetamine | Negative [N] | Negative | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Cannabinoids | Negative [N] | Negative | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Cocaine | Negative [N] | Negative | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Ecstasy | Negative [N] | Negative | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Methamphetamine | Negative [N] | Negative | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Opiate | Negative [N] | Negative | N |

Note 1: N=Normal, A=Different from reference value\_

Program: Listings\k345-lb-lst.sas



#### **Listing 16.2.8.1 - Individual laboratory measurements**

Category of Laboratory Parameters: VIROLOGY

| Subject<br>ID | Time<br>Point | Collection<br>Date/time | Parameter | Value and<br>Abnormality <sup>1</sup> | Normal Range or<br>Reference Value | Clinically<br>Significant? |
|---|---|---|---|---|---|---|
| S001/001 | Screening | ddMMMyyyy hh:mm | Hepatitis B Virus Surface Antigen | Negative [N] | Negative | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Hepatitis C Virus Antibody | Negative [N] | Negative | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | HIV Ag/Ab Combo | Negative [N] | Negative | N |
| ••• | | | <del></del> | | | ••• |

Note 1: N=Normal, A=Different from reference value

Program: Listings\k345-lb-lst.sas



#### Listing 16.2.8.1 - Individual laboratory measurements

## Category of Laboratory Parameters: ALCOHOL BREATH TEST AND PREGNANCY TEST

| Subject<br>ID | Time<br>Point | Collection<br>Date/time | Parameter | Value and<br>Abnormality <sup>1</sup> | Normal Range or<br>Reference Value | Clinically<br>Significant? |
|---|---|---|---|---|---|---|
| S001/001 | Screening | ddMMMyyyy hh:mm | Pregnancy Test | Negative [N] | Negative | N |
| S001/001 | Visit 2 - Day -1 | ddMMMyyyy hh:mm | Pregnancy Test | Negative [N] | Negative | N |
| S001/001 | Visit 2 - Day -1 | ddMMMyyyy hh:mm | Alcohol Breath Test | Negative [N] | Negative | N |
| S001/001 | Visit 4 - Day -1 | ddMMMyyyy hh:mm | Pregnancy Test | Negative [N] | Negative | N |
| S001/001 | Visit 4 - Day -1 | ddMMMyyyy hh:mm | Alcohol Breath Test | Negative [N] | Negative | N |
| | | | <del></del> | | | |

Note 1: N=Normal, A=Different from reference value\_

Program: Listings\k345-lb-lst.sas




#### **Listing 16.2.8.1 - Individual laboratory measurements**

# **Category of Laboratory Parameters: MICROBIOLOGICAL ANALYSIS**

| Subject<br>ID | Time<br>Point | Collection Date/time | Parameter | Value and<br>Abnormality <sup>1</sup> | Normal Range or<br>Reference Value | Clinically<br>Significant? |
|---|---|---|---|---|---|---|
| S001/001 | Visit 1.1 - Day -3/-2 | ddMMMyyyy hh:mm | Coronavirus SARS-COV-2 | Negative [N] | Negative | N |
| S001/001 | Visit 4 - Day -3/-2 | ddMMMyyyy hh:mm | Coronavirus SARS-COV-2 | Negative [N] | Negative | N |

Note 1: N=Normal, A=Different from reference value

Program: Listings\k345-lb-lst.sas



## Listing 16.2.8.2 - Investigator's interpretation of laboratory test results

| Subject<br>ID | Time<br>Point | Assessment<br>Date | Investigator's<br>Interpretation | Clinically<br>Significant<br>Abnormalites |
|---|---|---|---|---|
| S001/001 | Screening | ddMMMyyyy | Abnormal, Not Clinically Significant | |
| S001/001 | End of Study | ddMMMyyyy | Abnormal, Not Clinically Significant | |
| | ··· | | | |

Program: Listings\k345-lb-lst.sas



Listing 16.2.9.1 - Vital signs and body weight

| Subject<br>ID | Time<br>Point | Assessment Date/Time | Parameter | Value and<br>Abnormality <sup>1</sup> | Normal<br>Range | Clinically<br>Significant? |
|---|---|---|---|---|---|---|
| S001/001 | Screening | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 [N] | 60-89 | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 [N] | 50-90 | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Temperature [C] | 36.5 [N] | 35.7 - 37.5 | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Weight [kg] | 55.5 | | N |
| S001/001 | Visit 2 - Day -1 | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 | N |
| S001/001 | Visit 2 - Day -1 | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 [N] | 60-89 | N |
| S001/001 | Visit 2 - Day -1 | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 [N] | 50-90 | N |
| S001/001 | Visit 2 - Day -1 | ddMMMyyyy hh:mm | Temperature [C] | 36.5 [N] | 35.7 - 37.5 | N |
| S001/001 | Visit 3 - Day 1 - Pre-dose | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 | N |
| S001/001 | Visit 3 - Day 1 - Pre-dose | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 [N] | 60-89 | N |
| S001/001 | Visit 3 - Day 1 - Pre-dose | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 [N] | 50-90 | N |
| S001/001 | Visit 3 - Day 1 - Pre-dose | ddMMMyyyy hh:mm | Temperature [C] | 36.5 [N] | 35.7 - 37.5 | N |
| S001/001 | Visit 3 - Day 4 - 72 hour post-dose | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 | N |
| S001/001 | Visit 3 - Day 4 - 72 hour post-dose | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 [N] | 60-89 | N |
| S001/001 | Visit 3 - Day 4 - 72 hour post-dose | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 [N] | 50-90 | N |
| S001/001 | Visit 3 - Day 4 - 72 hour post-dose | ddMMMyyyy hh:mm | Temperature [C] | 36.5 [N] | 35.7 - 37.5 | N |
| S001/001 | Visit 5 - Day -1 | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 | N |
| S001/001 | Visit 5 - Day -1 | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 [N] | 60-89 | N |
| S001/001 | Visit 5 - Day -1 | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 [N] | 50-90 | N |
| S001/001 | Visit 5 - Day -1 | ddMMMyyyy hh:mm | Temperature [C] | 36.5 [N] | 35.7 - 37.5 | N |
| S001/001 | Visit 6 - Day 1 - Pre-dose | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 | N |
| S001/001 | Visit 6 - Day 1 - Pre-dose | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 [N] | 60-89 | N |
| S001/001 | Visit 6 - Day 1 - Pre-dose | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 [N] | 50-90 | N |
| S001/001 | Visit 6 - Day 1 - Pre-dose | ddMMMyyyy hh:mm | Temperature [C] | 36.5 [N] | 35.7 - 37.5 | N |

Note 1: N=Normal, H=Higher than upper normal limit, L=Lower than lower normal limit

Program: Listings\k345-vs-lst.sas



## Listing 16.2.9.1 - Vital signs and body weight

| Subject<br>ID | Time<br>Point | Assessment Date/Time | Parameter | Value and<br>Abnormality <sup>1</sup> | Normal<br>Range | Clinically<br>Significant? |
|---|---|---|---|---|---|---|
| S001/001 | Visit 6 - Day 4 - 72 hour post-dose | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 | N |
| S001/001 | Visit 6 - Day 4 - 72 hour post-dose | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 [N] | 60-89 | N |
| S001/001 | Visit 6 - Day 4 - 72 hour post-dose | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 [N] | 50-90 | N |
| S001/001 | Visit 6 - Day 4 - 72 hour post-dose | ddMMMyyyy hh:mm | Temperature [C] | 36.5 [N] | 35.7 - 37.5 | N |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Weight [kg] | 55.5 | | N |
| | | ••• | | | | |

Note 1: N=Normal, H=Higher than upper normal limit, L=Lower than lower normal limit

Program: Listings\k345-vs-lst.sas



## Listing 16.2.9.2 - Investigator's interpretation of ECG

| Subject<br>ID | Time<br>Point | Assessment<br>Date/Time | Investigator's<br>Interpretation |
|---|---|---|---|
| S001/001 | Screening | ddMMMyyyy hh:mm | Abnormal, Not Clinically Significant |
| S001/001 | Visit 2 - Day -1 | ddMMMyyyy hh:mm | Normal |
| S001/001 | Visit 3 - Day 1 - Pre-dose | ddMMMyyyy hh:mm | Normal |
| S001/001 | Visit 3 - Day 4 - 72 hour post-dose | ddMMMyyyy hh:mm | Abnormal, Not Clinically Significant |
| S001/001 | Visit 5 - Day -1 | ddMMMyyyy hh:mm | Normal |
| S001/001 | Visit 6 - Day 1 - Pre-dose | ddMMMyyyy hh:mm | Abnormal, Not Clinically Significant |
| S001/001 | Visit 6 - Day 4 - 72 hour post-dose | ddMMMyyyy hh:mm | Normal |

Program: Listings\k345-eg-lst.sas



## Listing 16.2.9.3 - Abnormal ECG parameters

| Subject<br>ID | Time<br>Point | Assessment Date/Time | Parameter | Value and Abnormality <sup>1</sup> | Clinically Significant? | If CS,<br>AE number |
|---|---|---|---|---|---|---|
| S001/001 | Screening | ddMMMyyyy hh:mm | Heart Rate [beats/min] | xx [L] | N | |
| S001/001 | Visit 3 - Day 4 - 72 hour post-dose | ddMMMyyyy hh:mm | QRS Duration [msec] | xx [H] | Y | 1 |
| S001/001 | Visit 3 - Day 4 - 72 hour post-dose | ddMMMyyyy hh:mm | QT Interval [msec] | xx [L] | N | |
| S001/001 | Visit 6 - Day 1 - Pre-dose | ddMMMyyyy hh:mm | QTcF Interval [msec] | xx [L] | N | |
| | | | | | ••• | |

Note 1: H=Higher than upper normal limit, L=Lower than lower normal limit

Program: Listings\k345-eg-lst.sas



## Listing 16.2.10.1 - Medical and surgical history

| Subject<br>ID | Category | Disease/Surgery<br>ID | | |
|---|---|---|---|---|
| S001/001 | Medical History | M1 | Verbatim: | Left shoulder luxation |
| | | | Preferred Term 1: | Joint dislocation |
| | | | System Organ Class 1: | Injury, poisoning and procedural complications |
| | | | Disease Start - End Date: | 2012 - 2012 |
| | Surgery | S1 | Verbatim: | Right knee meniscectomy |
| | | | Preferred Term 1: | Meniscus removal |
| | | | System Organ Class 1: | Surgical and medical procedures |
| | | | Surgery Date: | 04NOV1980 |
| | | ••• | | |

Note 1: MedDRA version 23.1 Program: Listings\k345-mh-lst.sas



## Listing 16.2.10.2 - Physical examination

| Subject<br>ID | Time Point | Physical<br>Examination<br>Date | | |
|---|---|---|---|---|
| S001/001 | Screening | ddMMMyyyy | Investigator's Interpretation | Normal |
| | Visit 3 - Day 4 - 72 hour post-dose | ddMMMyyyy | Investigator's Interpretation | Normal |
| | Visit 5 - Day -1 | ddMMMyyyy | Investigator's Interpretation | Normal |
| | End of Study | ddMMMyyyy | Investigator's Interpretation: | Abnormal, Clinically Significant |
| | | | Clinically Significant Abnormalities: | Left shoulder luxation |
| | | | Preferred Term 1: | Joint dislocation |
| | | | System Organ Class 1: | Injury, poisoning and procedural complications |
| ••• | | | | |

Note 1: MedDRA version 23.1 Program: Listings\k345-pe-lst.sas



## Listing 16.2.10.3 - Prior and concomitant medications

| Subject<br>ID | Category | Medication<br>ID | | |
|---|---|---|---|---|
| S001/001 | Prior | 1 | Verbatim: | Alerid |
| | | | Standardised Medication Name 1: | Alerid |
| | | | Active Ingredients 1: | Cetirizine hydrochloride |
| | | | Medication Class 1, 2: | Piperazine derivatives (R06AE) |
| | | | Indication: | Pollinosis |
| | | | Dose: | 10 mg |
| | | | Start - End Date/Time: | 2013 - Ongoing |
| | | | Frequency - Route: | 1 time per day - Oral |
| | | | Related to AE (AE nr.): | N (-) |
| | | | Related to MH (MH nr.): | Y (Disease M1) |
| | | | Related to SG (SG nr.): | N (-) |
| | Concomitant | 2 | Verbatim: | Paracen |
| | | | Standardised Medication Name 1: | Paracen |
| | | | Active Ingredients 1: | Paracetamol |
| | | | Medication Class <sup>1, 2</sup> : | Anilides (N02BE) |
| | | | Indication: | Headache |
| | | | Dose: | 500 mg |
| | | | Start - End Date/Time: | 15JUN2019 19:08 - 15JUN2019 19:08 |
| | | | Frequency - Route: | Once - Oral |
| | | | Related to AE (AE nr.): | Y (Adverse Event 1) |
| | | | Related to MH (MH nr.): | N (-) |
| | | | Related to SG (SG nr.): | N (-) |
| | ••• | ••• | | |

Note 1: WHO Drug Dictionary Enhanced March 1, 2020

Note 2: Anatomical Therapeutic Chemical classification, 4th level term

Program: Listings\k345-cm-lst.sas



Listing 16.2.10.4 - Subjects study visits

| Subject<br>ID | Visit | Visit Start Date (Day) | Visit End Date (Day) |
|---|---|---|---|
| S001/001 | Visit 1 - Screening - Day -21/-2 | ddMMMyyyy (-j) | |
| S001/001 | Visit 1.1 –Screening - Day -3/-2 | ddMMMyyyy (-y) | |
| S001/001 | Period 1 - Visit 2 - Day -1 | ddMMMyyyy (-1) | |
| S001/001 | Period 1 - Visit 3 - Days 1-4 | ddMMMyyyy (1) | ddMMMyyyy (4) |
| S001/001 | Period 2 - Visit 4 - Day -3/-2 | ddMMMyyyy (k-y) | |
| S001/001 | Period 2 - Visit 5 - Day -1 | ddMMMyyyy (k-1) | |
| S001/001 | Period 2 - Visit 6 - Days 1-4 | ddMMMyyyy (k+1) | ddMMMyyyy (k+4) |
| S001/001 | Final Visit | ddMMMyyyy (k+4) | |

Program: Listings\k345-sv-lst.sas



## Listing 16.2.10.5 - Fertility status and contraception

| Subject<br>ID | Chilbearing Potential? | Non-childbearing<br>Potential<br>Status Onset | Menopausal<br>Status? | Date of<br>Menopause | Surgical<br>Sterilisation? | Surgical<br>Sterilisation<br>Date | Reliable<br>Contraceptive<br>Method Used? |
|---|---|---|---|---|---|---|---|
| S001/001 | No | ddMMMyyyy | Yes | MMMyyyy | Yes | ddMMMyyyy | |
| ••• | | ••• | ••• | ••• | | ••• | ••• |

Note: Only female subjects are listed Program: Listings\k345-rp-lst.sas



#### **Listing 16.2.10.6 - Meals**

**Investigational Medicinal Product: Ladarixin fed (T)** 

| Subject<br>ID | Reference<br>Date/Time <sup>1</sup> | Meal<br>Nr | Standardised<br>Meal | Time Point | Meal<br>Served? | Meal Start<br>Date/time | Elapsed<br>Time | Fasting<br>Conditions<br>From 10 h<br>before<br>Breakfast? | Breakfast<br>completely<br>eaten<br>within<br>30 min? |
|---|---|---|---|---|---|---|---|---|---|
| S001/001 | ddMMMyyyy hh:mm | 1 | Breakfast | Day 1 –30 min before IMP admin | Y | ddMMMyyyy hh:mm | xx h xx min | Y | Y |
| S001/001 | ddMMMyyyy hh:mm | 2 | Lunch | Day 1 −5 hours post-dose | Y | ddMMMyyyy hh:mm | xx h xx min | | |
| S001/001 | ddMMMyyyy hh:mm | 3 | Dinner | Day 1 –12 hours post-dose | Y | ddMMMyyyy hh:mm | xx h xx min | | |
| S001/001 | | 4 | Breakfast | Day 2 –at about 09:00 | Y | ddMMMyyyy hh:mm | | | |
| S001/001 | | 5 | Lunch | Day 2 - at about 13:00 | Y | ddMMMyyyy hh:mm | | | |
| S001/001 | | 6 | Dinner | Day 2 - at about 20:00 | Y | ddMMMyyyy hh:mm | | | |
| S001/001 | | 7 | Breakfast | Day 3 - at about 09:00 | Y | ddMMMyyyy hh:mm | | | |
| S001/001 | | 8 | Lunch | Day 3 - at about 13:00 | Y | ddMMMyyyy hh:mm | | | |
| S001/001 | | 9 | Dinner | Day 3 - at about 20:00 | Y | ddMMMyyyy hh:mm | | | |

Note 1: Reference Date/time is Fasting conditions Start Date/Time for Day 1 – Breakfast (Test only) and IMP Administration Date/Time for Day 1 - Lunch and Day 1 - Dinner Note: Subjects are listed according to the product they actually received

Program: Listings\k345-ml-lst.sas



#### **Listing 16.2.10.6 - Meals**

**Investigational Medicinal Product: Ladarixin fasting (R)** 

| Subject<br>ID | Reference<br>Date/Time <sup>1</sup> | Meal<br>Nr | Standardised<br>Meal | Time Point | Meal<br>Served? | Meal Start<br>Date/time | Elapsed<br>Time | Fasting<br>Conditions<br>From 10 h<br>before<br>Breakfast? | Breakfast<br>completely<br>eaten<br>within<br>30 min? |
|---|---|---|---|---|---|---|---|---|---|
| S001/001 | ddMMMyyyy hh:mm | 11 | Lunch | Day 1 −5 hours post-dose | Y | ddMMMyyyy hh:mm | xx h xx min | | |
| S001/001 | ddMMMyyyy hh:mm | 12 | Dinner | Day 1 –12 hours post-dose | Y | ddMMMyyyy hh:mm | xx h xx min | | |
| S001/001 | | 13 | Breakfast | Day 2 –at about 09:00 | Y | ddMMMyyyy hh:mm | | | |
| S001/001 | | 14 | Lunch | Day 2 - at about 13:00 | Y | ddMMMyyyy hh:mm | | | |
| S001/001 | | 15 | Dinner | Day 2 - at about 20:00 | Y | ddMMMyyyy hh:mm | | | |
| S001/001 | | 16 | Breakfast | Day 3 - at about 09:00 | Y | ddMMMyyyy hh:mm | | | |
| S001/001 | | 17 | Lunch | Day 3 - at about 13:00 | Y | ddMMMyyyy hh:mm | | | |
| S001/001 | | 18 | Dinner | Day 3 - at about 20:00 | Y | ddMMMyyyy hh:mm | | | |
| | ••• | | | | | ••• | | | |

Note 1: Reference Date/time is Fasting conditions Start Date/Time for Day 1 - Breakfast (Test only) and IMP Administration Date/Time for Day 1 - Lunch and Day 1 - Dinner

Note: Subjects are listed according to the product they actually received

Program: Listings\k345-ml-lst.sas